CLINICAL TRIAL: NCT04886154
Title: A Phase I/II, Randomised, Controlled Study to Assess the Safety, Effectiveness and Immune Response of Meningococcal Combined ABCWY Vaccine When Administered to Healthy Adults (Phase I) and to Healthy Adolescents and Adults (Phase II)
Brief Title: A Study on the Safety, Effectiveness and Immune Response of Meningococcal Combined ABCWY Vaccine in Healthy Adolescents and Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 212458; 2020-004741-37 (EudraCT Number)
Record Dates: First submitted 2021-05-10; First posted 2021-05-13 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Infections, Meningococcal
Keywords: Bexsero; Menveo; Boostrix; MenABCWY-2Gen; Effectiveness; Safety; Invasive Meningococcal Disease; Adolescents and Adults
MeSH Terms: conditions — Meningococcal Infections | interventions — Vaccines; Saline Solution; 4CMenB vaccine; Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data will be collected in an observer-blind manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (15):
- ABCWY low dose Group (Experimental): Participants received two doses of the MenABCWY-2Gen low-dose vaccine on Day 1 and Day 31, following a 0, 1-month schedule during Study Phase I (Safety Lead-In).
  Interventions: Combination Product: MenABCWY-2Gen low dose vaccine
- Placebo low dose Group (Placebo Comparator): Participants received two doses of a placebo on Day 1 and Day 31, following a 0, 1-month schedule during Study Phase I (Safety Lead-In), as the control group for the ABCWY low-dose group.
  Interventions: Combination Product: Placebo
- ABCWY high dose Group (Experimental): Participants received two doses of the MenABCWY-2Gen high-dose vaccine on Day 1 and Day 31, following a 0, 1-month schedule during Study Phase I (Safety Lead-In).
  Interventions: Combination Product: MenABCWY-2Gen high dose vaccine
- Placebo high dose Group (Placebo Comparator): Participants received two doses of a placebo on Day 1 and Day 31, following a 0, 1-month schedule during Study Phase I (Safety Lead-In), as the control group for the ABCWY high-dose group.
  Interventions: Combination Product: Placebo
- ABCWY low dose_06 Group (Experimental): Participants received two doses of the MenABCWY-2Gen low-dose vaccine on Day 1 and Day 181, following a 0, 6-month schedule, along with one dose of a placebo on Day 121 during Phase II (Formulation and Schedule-Finding).
  Interventions: Combination Product: MenABCWY-2Gen low dose vaccine; Combination Product: Placebo
- ABCWY low dose_02 Group (Experimental): Participants received two doses of the MenABCWY-2Gen low-dose vaccine on Day 121 and Day 181, following a 0, 2-month schedule, along with one dose of a placebo on Day 1 during Phase II (Formulation and Schedule-Finding).
  Interventions: Combination Product: MenABCWY-2Gen low dose vaccine; Combination Product: Placebo
- ABCWY high dose_06 Group (Experimental): Participants received two doses of the MenABCWY-2Gen high-dose vaccine on Day 1 and Day 181, following a 0, 6-month schedule, along with one dose of a placebo on Day 121 during Phase II (Formulation and Schedule-Finding).
  Interventions: Combination Product: MenABCWY-2Gen high dose vaccine; Combination Product: Placebo
- ABCWY high dose_02 Group (Experimental): Participants received two doses of the MenABCWY-2Gen high-dose vaccine on Day 121 and Day 181, following a 0, 2-month schedule, along with one dose of a placebo on Day 1 during Phase II (Formulation and Schedule-Finding).
  Interventions: Combination Product: MenABCWY-2Gen high dose vaccine; Combination Product: Placebo
- Control Group (Active Comparator): Participants randomized to the control group received two doses of the Bexsero (MenB) vaccine on Day 1 and Day 181, following a 0, 6-month schedule, and one dose of Menveo (MenACWY) on Day 1 during Study Phase II (Formulation and Schedule-Finding).
  Interventions: Combination Product: MenB vaccine; Biological: MenACWY vaccine
- ABCWY low dose_01 Group (Experimental): Participants received two doses of MenABCWY-2Gen low dose vaccine on Day 1 and Day 31, following a 0, 1-month schedule during study Phase II (Sourcing).
  Interventions: Combination Product: MenABCWY-2Gen low dose vaccine
- ABCWY high dose_01 Group (Experimental): Participants received two doses of MenABCWY-2Gen high dose vaccine on Day 1 and Day 31, following a 0, 1-month schedule during study Phase II (Sourcing).
  Interventions: Combination Product: MenABCWY-2Gen high dose vaccine
- ABCWY low doseS_02 Group (Experimental): Participants received two doses of MenABCWY-2Gen low dose vaccine on Day 1 and day 61 following a 0, 2-month schedule during study Phase II (Sourcing).
  Interventions: Combination Product: MenABCWY-2Gen low dose vaccine
- ABCWY high doseS_02 Group (Experimental): Participants received two doses of MenABCWY-2Gen high dose vaccine on Day 1 and day 61 following a 0, 2-month schedule during study Phase II (Sourcing).
  Interventions: Combination Product: MenABCWY-2Gen high dose vaccine
- ABCWY low doseS_06 Group (Experimental): Participants received two doses of MenABCWY-2Gen low dose vaccine on Day 1 and day 181 following a 0, 6-month schedule during study Phase II (Sourcing).
  Interventions: Combination Product: MenABCWY-2Gen low dose vaccine
- ABCWY high doseS_06 Group (Experimental): Participants received two doses of MenABCWY-2Gen high dose vaccine on Day 1 and day 181 following a 0, 6-month schedule during study Phase II (Sourcing).
  Interventions: Combination Product: MenABCWY-2Gen high dose vaccine

INTERVENTIONS:
Combination Product: MenABCWY-2Gen low dose vaccine — MenABCWY-2Gen low dose vaccine is administered intramuscularly as 2 doses to participants in the ABCWY low dose Group in study Phase I, ABCWY low dose_06 Group and ABCWY low dose_02 Group in study Phase II (Formulation and Schedule-finding) and as 2 doses to participants in the ABCWY low dose_01 Group, ABCWY low doseS_02 Group and ABCWY low doseS_06 Group in study Phase II (Sourcing).
  Arms: ABCWY low dose Group; ABCWY low doseS_02 Group; ABCWY low doseS_06 Group; ABCWY low dose_01 Group; ABCWY low dose_02 Group; ABCWY low dose_06 Group
Combination Product: MenABCWY-2Gen high dose vaccine — MenABCWY-2Gen high dose vaccine is administered intramuscularly 2 doses to participants in the ABCWY high dose Group in study Phase I, ABCWY high dose_06 Group and ABCWY high dose_02 Group in study Phase II (Formulation and Schedule-finding) and as 2 doses to participants in the ABCWY high dose_01 Group, ABCWY high doseS_02 Group and ABCWY high doseS_06 Group in study Phase II (Sourcing).
  Arms: ABCWY high dose Group; ABCWY high doseS_02 Group; ABCWY high doseS_06 Group; ABCWY high dose_01 Group; ABCWY high dose_02 Group; ABCWY high dose_06 Group
Combination Product: Placebo — Placebo is administered intramuscularly as 2 doses to participants in the Placebo low dose Group, Placebo high dose Group in study Phase I and as 1 dose to participants in the ABCWY low dose_06 Group, ABCWY low dose_02 Group, ABCWY high dose_06 Group, ABCWY high dose_02 Group in study Phase II (Formulation and Schedule-finding).
  Other Names: NaCl, saline solution
  Arms: ABCWY high dose_02 Group; ABCWY high dose_06 Group; ABCWY low dose_02 Group; ABCWY low dose_06 Group; Placebo high dose Group; Placebo low dose Group
Combination Product: MenB vaccine — MenB vaccine is administered intramuscularly as 2 doses in a 0,6-months schedule to participants in the Control Group in study Phase II (Formulation and Schedule-finding).
  Other Names: GSK's meningococcal group B vaccine, Bexsero
  Arms: Control Group
Biological: MenACWY vaccine — MenACWY vaccine is administered intramuscularly as 1 dose to participants in the Control Group in study Phase II (Formulation and Schedule-finding).
  Other Names: GSK's combined meningococcal groups A, C, Y and W-135 conjugate vaccine, Menveo
  Arms: Control Group

SUMMARY:
The purpose of this study was to assess the safety, effectiveness, and immune response of the meningococcal combined ABCWY vaccine (GSK4023393A) intended to protect against invasive meningococcal disease (IMD) caused by all 5 meningococcal serogroups. The first time-in-human (FTIH), Phase I part of this study was conducted in healthy adults in a dose-escalating fashion with 2 formulations of the investigational MenABCWY-2Gen vaccine and served as a safety lead-in to the Phase II study. The Phase II part of the study was conducted in 2 parts: The 'formulation and schedule-finding' part followed in healthy adolescents and young adults and was designed to select the vaccine formulation and the schedule to be tested in Phase III. The 'blood sourcing' part was conducted in healthy adults in order to collect sufficient serum samples for the development of assays to be used in the MenABCWY-2Gen vaccine clinical development program.

ELIGIBILITY:
Inclusion Criteria:

All inclusion criteria are applicable for both study phases, except where specified otherwise.

* Participants and/or participants' parent(s)/Legally Acceptable Representative(s) (LAR) who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g. completion of the eDiaries, return for follow-up visits).
* Written or witnessed/thumb printed informed consent obtained from the participant or /parent(s)/LAR(s) of the participant prior to performance of any study specific procedure.
* Written informed assent obtained from the participant (if applicable) prior to performing any study specific procedure.
* Phase I only: A male or female between, and including, 18 and 40 years of age (i.e. 40 years + 364 days) at the time of the first study intervention administration.
* Phase II (Formulation and Schedule-finding) only: A male or female between, and including, 10 and 25 years of age (i.e. 25 years + 364 days) at the time of the first study intervention administration.
* Phase II (Sourcing) only: A male or female between, and including, 18 and 50 years of age (i.e. 50 years + 364 days) at the time of the first study intervention administration.
* Participants who are either unvaccinated with MenACWY vaccine or have received a single previous dose of MenACWY vaccine can participate in the study, if they have received it at least 4 years prior to informed consent and assent as applicable (with the exception of meningococcal C vaccination, if the last dose of MenC was received at ≤24 months of age).
* Healthy participants as established by medical history and clinical examination before entering into the study.
* Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause.
* Female participants of childbearing potential may be enrolled in the study, if the participant:

  * has practiced adequate contraception for 1 month prior to study intervention administration, and
  * has a negative pregnancy test on the day of study intervention administration, and
  * has agreed to continue adequate contraception during the entire treatment period and for 1 month after completion of the study intervention administration.

Exclusion Criteria:

Medical conditions

* Current or previous, confirmed or suspected disease caused by N. meningitidis.
* Household contact with and/or intimate exposure to an individual with laboratory confirmed N. meningitidis infection within 60 days of enrolment.
* Progressive, unstable or uncontrolled clinical conditions.
* Clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
* Are obese at enrolment (e.g. for participants from 20 years of age a body mass index (BMI) ≥ 30 kg/m2, for participants up to 19 years of age a BMI ≥ 95th percentile for age and gender or as applicable per country recommendations).
* Any neuroinflammatory (including but not limited to: demyelinating disorders, encephalitis or myelitis of any origin), congenital neurological conditions, encephalopathies, seizures (including all subtypes such as: absence seizures, generalised tonic-clonic seizures, partial complex seizures, partial simple seizures). History of febrile convulsions should not lead to exclusion.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study interventions.
* Hypersensitivity, including allergy, to any component of vaccines, including diphtheria toxoid (CRM197) and latex medicinal products or medical equipment whose use is foreseen in this study.
* Abnormal function or modification of the immune system resulting from:

  * Autoimmune disorders (including, but not limited to: blood, endocrine, hepatic, muscular, nervous system or skin autoimmune disorders; lupus erythematosus and associated conditions; rheumatoid arthritis and associated conditions; scleroderma and associated disorders) or immunodeficiency syndromes (including, but not limited to: acquired immunodeficiency syndromes and primary immunodeficiency syndromes).
  * Systemic administration of corticosteroids (PO/IV/IM) for more than 14 consecutive days within 3 months prior to study vaccination until the last blood sampling visit for Phase I and Phase II (Sourcing) and Visit 5 (Day 211) for Phase II (Formulation and Schedule-finding). This will mean prednisone equivalent ≥20 mg/day for adult participants/ ≥0.5 mg/kg/day with maximum of 20 mg/day for paediatric participants. Inhaled and topical steroids are allowed.
  * Administration of antineoplastic and immunomodulating agents or radiotherapy within 90 days prior to study vaccination.
  * Administration of long-acting immune-modifying drugs at any time during the study period (e.g. infliximab).
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.

Prior/Concomitant therapy

* Use of any investigational or non-registered product (drug, vaccine or medical device) other than the study intervention(s) during the period beginning 30 days before the first dose of study intervention(s) (Day -29 to Day 1), or their planned use during the study period.
* Previous vaccination against any group B meningococcal vaccine at any time prior to informed consent and assent as applicable.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 3 months before the administration of the first dose of study intervention(s) or planned administration until the last blood sampling visit for Phase I and Phase II (Sourcing) and Visit 5 (Day 211) for Phase II (Formulation and Schedule-finding).
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 3 months prior to the first study intervention dose(s) until the last blood sampling visit for Phase I and Phase II (Sourcing) and Visit 5 (Day 211) for Phase II (Formulation and Schedule-finding). For corticosteroids, this will mean prednisone equivalent ≥20 mg/day for adult participants/ ≥0.5 mg/kg/day with maximum of 20 mg/day for paediatric participants. Inhaled and topical steroids are allowed.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug/invasive medical device).

Other exclusions

* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* History of /current chronic alcohol abuse and/or drug abuse as determined by the investigator.
* Any study personnel or immediate dependents, family, or household member.
* Phase II (Formulation and Schedule-finding): Child in care.

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1440 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (46):
- United States (12):
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Longmont, Colorado
  - GSK Investigational Site, Doral, Florida
  - GSK Investigational Site, Miami Lakes, Florida
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, San Antonio, Texas
- Australia (6):
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Fortitude Valley, Queensland
  - GSK Investigational Site, Taringa, Queensland
  - GSK Investigational Site, Tarragindi, Queensland
  - GSK Investigational Site, Nedlands, Western Australia
  - GSK Investigational Site, Spearwood, Western Australia
- Belgium (4):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Linkebeek
- Brazil (4):
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, Salvador
  - GSK Investigational Site, São José do Rio Preto
  - GSK Investigational Site, São Paulo
- Finland (2):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Turku
- Poland (11):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Luboń
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Tarnów
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Trzebnica
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Sweden (5):
  - GSK Investigational Site, Borås
  - GSK Investigational Site, Karlskrona
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Umeå
- Turkey (Türkiye) (2):
  - GSK Investigational Site, Istanbul
  - GSK Investigational Site, Kocaeli

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 1440 participants enrolled, 3 participants from Phase II (Formulation and Schedule-finding) did not receive vaccination as they did not meet the eligibility criteria, therefore only 1437 participants were included in the Exposed Set and started the study.
Period: Overall Study
Arm/Group | ABCWY Low Dose Group | Placebo Low Dose Group | ABCWY High Dose Group | Placebo High Dose Group | ABCWY Low dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_06 Group | ABCWY High dose_02 Group | Control Group | ABCWY Low dose_01 Group | ABCWY High dose_01 Group | ABCWY Low doseS_02 Group | ABCWY High doseS_02 Group | ABCWY Low doseS_06 Group | ABCWY High doseS_06 Group
Started | 12 | 4 | 13 | 3 | 239 | 181 | 238 | 194 | 197 | 54 | 53 | 62 | 62 | 62 | 63
Completed | 11 | 4 | 11 | 3 | 209 | 166 | 218 | 175 | 182 | 53 | 50 | 59 | 61 | 60 | 56
Not Completed | 1 | 0 | 2 | 0 | 30 | 15 | 20 | 19 | 15 | 1 | 3 | 3 | 1 | 2 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 3
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0 | 17 | 7 | 8 | 7 | 8 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — ADVERSE EVENT REQUIRING EXPEDITED REPORT | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — MIGRATED / MOVED FROM THE STUDY AREA | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other, Not Specified | 0 | 0 | 0 | 0 | 11 | 8 | 9 | 10 | 6 | 1 | 1 | 2 | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABCWY Low Dose Group | Placebo Low Dose Group | ABCWY High Dose Group | Placebo High Dose Group | ABCWY Low dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_06 Group | ABCWY High dose_02 Group | Control Group | ABCWY Low dose_01 Group | ABCWY High dose_01 Group | ABCWY Low doseS_02 Group | ABCWY High doseS_02 Group | ABCWY Low doseS_06 Group | ABCWY High doseS_06 Group | Total
Number analyzed (Participants) | 12 | 4 | 13 | 3 | 239 | 181 | 238 | 194 | 197 | 54 | 53 | 62 | 62 | 62 | 63 | 1437
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (7.5) | 30.8 (6.2) | 31.7 (6.0) | 28.7 (3.8) | 18.9 (4.7) | 18.6 (4.6) | 18.7 (5.0) | 18.6 (4.7) | 18.4 (4.6) | 34.6 (8.9) | 31.7 (7.3) | 35.2 (9.1) | 34.6 (8.4) | 37.0 (8.7) | 37.3 (8.8) | 23.0 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 7 | 1 | 153 | 96 | 156 | 121 | 113 | 28 | 34 | 38 | 39 | 37 | 37 | 868
  Male | 6 | 2 | 6 | 2 | 86 | 85 | 82 | 73 | 84 | 26 | 19 | 24 | 23 | 25 | 26 | 569
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 41 | 29 | 30 | 29 | 35 | 3 | 6 | 0 | 0 | 3 | 0 | 176
  Not Hispanic or Latino | 11 | 4 | 13 | 3 | 198 | 152 | 208 | 165 | 162 | 50 | 46 | 62 | 62 | 59 | 63 | 1258
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Administration Site Events in Study Phase I (Safety Lead-in)
Description: The solicited administration site events include injection site pain, erythema (redness), swelling and induration. Any solicited administration site AEs = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 7 days (including the day of vaccination) following vaccination at Day 1
Population: Analysis was performed on the Phase I Exposed set (ES), which included all participants who received at least one dose of the study treatment and have post-vaccination data for the specified analysis at specified timepoints. Allocation per group using the enrolled set is based on the treatment administered.
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low Dose Group | Placebo Low Dose Group | ABCWY High Dose Group | Placebo High Dose Group
Number analyzed (Participants) | 12 | 4 | 13 | 3
Participants
  Erythema | 0 | 0 | 0 | 0
  Induration | 1 | 0 | 0 | 0
  Pain | 11 | 1 | 13 | 0
  Swelling | 1 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Solicited Administration Site Events in Study Phase I (Safety Lead-in)
Description: as for outcome 1
Time Frame: During the 7 days (including the day of vaccination) following vaccination at Day 31
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low Dose Group | Placebo Low Dose Group | ABCWY High Dose Group | Placebo High Dose Group
Number analyzed (Participants) | 12 | 4 | 11 | 3
Participants
  Erythema | 2 | 0 | 0 | 0
  Induration | 0 | 0 | 0 | 0
  Pain | 8 | 1 | 8 | 1
  Swelling | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Solicited Systemic Events in Study Phase I (Safety Lead-in)
Description: The solicited systemic events include fever (temperature ≥ 38.0°C), nausea, fatigue, myalgia, arthralgia and headache.
Time Frame: During the 7 days (including the day of vaccination) following vaccination at Day 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low Dose Group | Placebo Low Dose Group | ABCWY High Dose Group | Placebo High Dose Group
Number analyzed (Participants) | 12 | 4 | 13 | 3
Participants
  Arthralgia | 1 | 1 | 2 | 1
  Fatigue | 4 | 1 | 11 | 2
  Headache | 4 | 0 | 4 | 1
  Myalgia | 4 | 0 | 3 | 1
  Nausea | 0 | 0 | 3 | 0
  Fever (C) | 1 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Solicited Systemic Events in Study Phase I (Safety Lead-in)
Description: The solicited systemic events include fever (temperature ≥ 38.0°C), nausea, fatigue, myalgia, arthralgia and headache.
Time Frame: During the 7 days (including the day of vaccination) following vaccination at Day 31
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low Dose Group | Placebo Low Dose Group | ABCWY High Dose Group | Placebo High Dose Group
Number analyzed (Participants) | 12 | 4 | 11 | 3
Participants
  Arthralgia | 1 | 2 | 2 | 0
  Fatigue | 1 | 2 | 7 | 2
  Headache | 4 | 2 | 3 | 1
  Myalgia | 1 | 1 | 2 | 0
  Nausea | 1 | 1 | 2 | 0
  Fever (C) | 1 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Any Unsolicited Adverse Events (AEs), Including All Serious Adverse Events (SAEs), AEs Leading to Withdrawal and AEs of Special Interest (AESIs) in Study Phase I (Safety Lead-in)
Description: Unsolicited AEs includes any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is reported as an unsolicited adverse event. A SAE is any untoward medical occurrence that results in death, is life-threatening, requires or prolongs hospitalization, results in disability/incapacity and is a congenital anomaly/birth defect in a subject's offspring. AESIs are predefined (serious or non-serious) AEs of scientific and medical concern specific to the product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor can be appropriate, because such an event might warrant further investigation to characterize and understand it. A participant was considered withdrawn if no study procedures occurred, and no follow-up or further information has been collected from the date of withdrawal or last contact.
Time Frame: During the 30 days (including the day of vaccination) following vaccination at Day 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low Dose Group | Placebo Low Dose Group | ABCWY High Dose Group | Placebo High Dose Group
Number analyzed (Participants) | 12 | 4 | 13 | 3
Participants | 4 | 1 | 8 | 1

6. Primary Outcome: Number of Participants With Any Unsolicited AEs, Including All SAEs, AEs Leading to Withdrawal and AESIs in Study Phase I (Safety Lead-in)
Description: as for outcome 5
Time Frame: During the 30 days (including the day of vaccination) following vaccination at Day 31
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low Dose Group | Placebo Low Dose Group | ABCWY High Dose Group | Placebo High Dose Group
Number analyzed (Participants) | 12 | 4 | 11 | 3
Participants | 6 | 1 | 7 | 0

7. Primary Outcome: Number of Participants With SAEs, AEs Leading to Withdrawal and AESIs in Study Phase I (Safety Lead-in)
Description: A SAEs is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity and is a congenital anomaly/birth defect in the offspring of a study subject. AESIs are predefined (serious or non-serious) AEs of scientific and medical concern specific to the product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor can be appropriate, because such an event might warrant further investigation to characterize and understand it. A participant was considered withdrawn if no study procedures occurred, and no follow-up or further information has been collected from the date of withdrawal or last contact.
Time Frame: Throughout the Phase 1 study period (Day 1 through Day 211)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low Dose Group | Placebo Low Dose Group | ABCWY High Dose Group | Placebo High Dose Group
Number analyzed (Participants) | 12 | 4 | 13 | 3
Participants
  SAEs | 0 | 0 | 0 | 0
  AEs leading to withdrawal | 0 | 0 | 0 | 0
  AESIs | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Change From Baseline in Haematological and Biochemical Laboratory Values, in Study Phase I (Safety Lead-in)
Description: The safety laboratory data included haematological parameters (basophils, eosinophils, Erythrocytes, hemoglobin, leukocytes, lymphocytes, monocytes, platelets and neutrophils), and chemical parameters (Alanine Aminotransferase [ALT], Aspartate Aminotransferase [AST], Creatinine) Below = value below the laboratory reference range defined for the specified visit and laboratory parameter; Within = value within the laboratory reference range defined for the specified visit and laboratory parameter; Above = value above the laboratory reference range defined for the specified visit and laboratory parameter.
Time Frame: At Day 8 (7 days after the first vaccination)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low Dose Group | Placebo Low Dose Group | ABCWY High Dose Group | Placebo High Dose Group
Number analyzed (Participants) | 12 | 4 | 13 | 3
Participants
  Basophils: Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Basophils: Within (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Basophils: Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Basophils: Below (baseline) - within (Day 8) | 0 | 0 | 0 | 0
  Basophils: Within (baseline) - within (Day 8) | 12 | 4 | 13 | 3
  Basophils: Above (baseline) - within (Day 8) | 0 | 0 | 0 | 0
  Basophils: Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Basophils: WIthin (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Basophils: Above (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Eosinophils: Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Eosinophils: Within (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Eosinophils: Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Eosinophils: Below (baseline) - within (Day 8) | 0 | 0 | 0 | 0
  Eosinophils: Within (baseline) - within (Day 8) | 11 | 4 | 13 | 3
  Eosinophils: Above (baseline) - within (Day 8) | 0 | 0 | 0 | 0
  Eosinophils: Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Eosinophils: WIthin (baseline) - above (Day 8) | 1 | 0 | 0 | 0
  Eosinophils: Above (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Erythrocytes: Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Erythrocytes: Within (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Erythrocytes: Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Erythrocytes: Below (baseline) - within (Day 8) | 0 | 0 | 1 | 0
  Erythrocytes: Within (baseline) - within (Day 8) | 12 | 4 | 12 | 3
  Erythrocytes: Above (baseline) - within (Day 8) | 0 | 0 | 0 | 0
  Erythrocytes: Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Erythrocytes: WIthin (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Erythrocytes: Above (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Hemoglobin: Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Hemoglobin: Within (baseline) - below (Day 8) | 0 | 0 | 2 | 0
  Hemoglobin: Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Hemoglobin: Below (baseline) - within (Day 8) | 0 | 0 | 0 | 0
  Hemoglobin: Within (baseline) - within (Day 8) | 12 | 4 | 11 | 3
  Hemoglobin: Above (baseline) - within (Day 8) | 0 | 0 | 0 | 0
  Hemoglobin: Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Hemoglobin: WIthin (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Hemoglobin: Above (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Leukocytes: Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Leukocytes: Within (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Leukocytes: Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Leukocytes: Below (baseline) - within (Day 8) | 0 | 0 | 0 | 0
  Leukocytes: Within (baseline) - within (Day 8) | 12 | 4 | 13 | 3
  Leukocytes: Above (baseline) - within (Day 8) | 0 | 0 | 0 | 0
  Leukocytes: Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Leukocytes: WIthin (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Leukocytes: Above (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Lymphocytes: Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Lymphocytes: Within (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Lymphocytes: Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Lymphocytes: Below (baseline) - within (Day 8) | 0 | 0 | 0 | 0
  Lymphocytes: Within (baseline) - within (Day 8) | 12 | 4 | 13 | 3
  Lymphocytes: Above (baseline) - within (Day 8) | 0 | 0 | 0 | 0
  Lymphocytes: Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Lymphocytes: WIthin (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Lymphocytes: Above (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Monocytes: Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Monocytes: Within (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Monocytes: Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Monocytes: Below (baseline) - within (Day 8) | 0 | 0 | 0 | 0
  Monocytes: Within (baseline) - within (Day 8) | 12 | 4 | 13 | 3
  Monocytes: Above (baseline) - within (Day 8) | 0 | 0 | 0 | 0
  Monocytes: Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Monocytes: WIthin (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Monocytes: Above (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Neutrophils: Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Neutrophils: Within (baseline) - below (Day 8) | 0 | 1 | 0 | 0
  Neutrophils: Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Neutrophils: Below (baseline) - within (Day 8) | 0 | 0 | 1 | 0
  Neutrophils: Within (baseline) - within (Day 8) | 12 | 3 | 12 | 3
  Neutrophils: Above (baseline) - within (Day 8) | 0 | 0 | 0 | 0
  Neutrophils: Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Neutrophils: WIthin (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Neutrophils: Above (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Platelets: Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Platelets: Within (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Platelets: Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Platelets: Below (baseline) - within (Day 8) | 1 | 0 | 1 | 0
  Platelets: Within (baseline) - within (Day 8) | 11 | 4 | 12 | 3
  Platelets: Above (baseline) - within (Day 8) | 0 | 0 | 0 | 0
  Platelets: Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Platelets: WIthin (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Platelets: Above (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Alanine Aminotransferase (ALT): Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Alanine Aminotransferase (ALT): Within (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Alanine Aminotransferase (ALT): Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Alanine Aminotransferase (ALT): Below (baseline) - within (Day 8) | 0 | 0 | 0 | 0
  Alanine Aminotransferase (ALT): Within (baseline) - within (Day 8) | 10 | 4 | 10 | 2
  Alanine Aminotransferase (ALT): Above (baseline) - within (Day 8) | 1 | 0 | 0 | 0
  Alanine Aminotransferase (ALT): Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Alanine Aminotransferase (ALT): WIthin (baseline) - above (Day 8) | 0 | 0 | 1 | 1
  Alanine Aminotransferase (ALT): Above (baseline) - above (Day 8) | 1 | 0 | 2 | 0
  Aspartate Aminotransferase (AST): Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Aspartate Aminotransferase (AST): Within (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Aspartate Aminotransferase (AST): Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Aspartate Aminotransferase (AST): Below (baseline) - within (Day 8) | 0 | 0 | 0 | 0
  Aspartate Aminotransferase (AST): Within (baseline) - within (Day 8) | 12 | 4 | 12 | 2
  Aspartate Aminotransferase (AST): Above (baseline) - within (Day 8) | 0 | 0 | 0 | 0
  Aspartate Aminotransferase (AST): Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Aspartate Aminotransferase (AST): WIthin (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Aspartate Aminotransferase (AST): Above (baseline) - above (Day 8) | 0 | 0 | 1 | 1
  Creatinine: Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Creatinine: Within (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Creatinine: Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0
  Creatinine: Below (baseline) - within (Day 8) | 0 | 0 | 1 | 0
  Creatinine: Within (baseline) - within (Day 8) | 12 | 3 | 12 | 2
  Creatinine: Above (baseline) - within (Day 8) | 0 | 1 | 0 | 1
  Creatinine: Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Creatinine: WIthin (baseline) - above (Day 8) | 0 | 0 | 0 | 0
  Creatinine: Above (baseline) - above (Day 8) | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Clinically Significant Haematological and Biochemical Laboratory Values, in Study Phase I (Safety Lead-in)
Description: Clinical laboratory testing included hematological and biochemical laboratory values. Any abnormal laboratory test result (e.g., in hematology or clinical chemistry) that was deemed clinically significant by the investigator's medical and scientific judgment, and not related to an underlying disease, was reported as an unsolicited adverse event (AE) unless it was considered by the investigator to be more severe than expected for the participant's condition. The safety laboratory data included hematological parameters (basophils, eosinophils, erythrocytes, hemoglobin, leukocytes, lymphocytes, monocytes, platelets, and neutrophils) and chemical parameters (Alanine Aminotransferase [ALT], Aspartate Aminotransferase [AST], and creatinine).
Time Frame: At Day 8 (7 days after the first vaccination)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low Dose Group | Placebo Low Dose Group | ABCWY High Dose Group | Placebo High Dose Group
Number analyzed (Participants) | 12 | 4 | 13 | 3
Participants
  Basophils | 0 | 0 | 0 | 0
  Eosinophils | 0 | 0 | 0 | 0
  Erythrocytes | 0 | 0 | 0 | 0
  Hemoglobin | 0 | 0 | 0 | 0
  Leukocytes | 0 | 0 | 0 | 0
  Lymphocytes | 0 | 0 | 0 | 0
  Monocytes | 0 | 0 | 0 | 0
  Neutrophils | 0 | 0 | 0 | 0
  Platelets | 0 | 0 | 0 | 0
  Alanine Aminotransferase (ALT) | 0 | 0 | 0 | 0
  Aspartate Aminotransferase (AST) | 0 | 0 | 0 | 0
  Creatinine | 0 | 0 | 0 | 0

10. Primary Outcome: Percentage of Blood Samples With Bactericidal Serum Activity Using Enc-hSBA Against a Panel of 110 Randomly Selected Endemic US N. Meningitidis Serogroup B Invasive Disease Strains at Study Phase II (Formulation and Schedule-finding)
Description: The effectiveness of the MenABCWY-2Gen (low & high dose) vaccine when administered at 0,2- or 0,6-months schedule compared to MenB vaccine administered at 0,6-months schedule, against a panel of 110 randomly selected endemic N. meningitidis serogroup B strains is measured in terms of percentage of samples with bactericidal activity using endogenous complement human Serum Bactericidal Assay (enc-hSBA), which provides a qualitative assessment (yes/no) of the presence of sufficient bactericidal antibodies in human sera to kill a meningococcal strain at a specific dilution of 1:4.
Time Frame: At Day 211 (1 month after the last vaccination)
Population: Analysis was performed on the Phase II Formulation and Schedule-finding (FSF) Full Analysis Set (FAS), which included all participants who received at least one dose of the study treatment and have post-vaccination immunogenicity data for the specified analysis at specified timepoints. The allocation in a group is done in function of the randomised treatment.
  Number of Participants analyzed = Total number of participants included in FAS.
Measure: Number; unit: Percentage of blood Samples
Units Other Than Participants: Samples
Arm/Group | ABCWY Low dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_06 Group | ABCWY High dose_02 Group | Control Group
Number analyzed (Participants) | 230 | 177 | 235 | 189 | 194
Number analyzed (Samples) | 6714 | 5383 | 7063 | 5540 | 5620
Percentage of blood Samples | 91.0 | 86.2 | 91.0 | 88.4 | 86.4
Statistical Analysis 1: Comparison: ABCWY Low dose_06 Group vs Control Group; To demonstrate the superiority of the effectiveness of the MenABCWY-2Gen vaccine (low dose) when administered at 0,6-months schedule, compared to the MenB vaccine administered at 0,6-months schedule; Test type: Superiority — Superiority was to be demonstrated if the lower limit of the 2-sided 97.5% CI for the difference in percentages of samples with bactericidal serum activity is above 5% between the ABCWY low dose_06 group compared to the Control group at 1 month after the last vaccination; Difference in percentage = 4.67, 97.5% CI 2-sided [3.38 to 5.97] — The 97.5% CIs for the difference in percentages between ABCWY low dose_06 group and the control group is constructed using the method of Miettinen and Nurminen
Statistical Analysis 2: Comparison: ABCWY Low dose_02 Group vs Control Group; To demonstrate the superiority of the effectiveness of the MenABCWY-2Gen vaccine (low dose) when administered at 0,2- months schedule, compared to the MenB vaccine administered at 0,6-months schedule; Test type: Superiority — Superiority was to be demonstrated if the lower limit of the 2-sided 97.5% CI for the difference in percentages of samples with bactericidal serum activity is above 5% between the ABCWY low dose_02 group compared to the Control group at 1 month after the last vaccination; Difference in percentage = -0.17, 97.5% CI 2-sided [-1.65 to 1.30] — The 97.5% CIs for the difference in percentages between ABCWY low dose_02 group and the control group is constructed using the method of Miettinen and Nurminen
Statistical Analysis 3: Comparison: ABCWY High dose_06 Group vs Control Group; To demonstrate the superiority of the effectiveness of the MenABCWY-2Gen vaccine (high dose) when administered at 0,6- months schedule, compared to the MenB vaccine administered at 0,6-months schedule; Test type: Superiority — Superiority was to be demonstrated if the lower limit of the 2-sided 97.5% CI for the difference in percentages of samples with bactericidal serum activity is above 5% between the ABCWY high dose_06 group compared to the Control group at 1 month after the last vaccination; Difference in percentage = 4.60, 97.5% CI 2-sided [3.33 to 5.89] — The 97.5% CIs for the difference in percentages between ABCWY high dose_06 group and the control group is constructed using the method of Miettinen and Nurminen
Statistical Analysis 4: Comparison: ABCWY High dose_02 Group vs Control Group; To demonstrate the superiority of the effectiveness of the MenABCWY-2Gen vaccine (high dose) when administered at 0,2- months schedule, compared to the MenB vaccine administered at 0,6-months schedule; Test type: Superiority — Superiority was to be demonstrated if the lower limit of the 2-sided 97.5% CI for the difference in percentages of samples with bactericidal serum activity is above 5% between the ABCWY high dose_02 group compared to the Control group at 1 month after the last vaccination; Difference in percentage = 2.01, 97.5% CI 2-sided [0.60 to 3.42] — The 97.5% CIs for the difference in percentages between ABCWY high dose_02 group and the control group is constructed using the method of Miettinen and Nurminen

11. Primary Outcome: Number of Participants With a 4-fold Rise in hSBA Titers Against Serogroups A, C, W and Y in Study Phase II (Formulation and Schedule-finding)
Description: The immune response to the MenABCWY-2Gen (low and high dose) vaccine when administered at 0,2- or 0,6-months schedule compared to MenACWY vaccine (single dose), relative to day 1 in the ABCWY and control groups (0, 6 month schedule) and day 31 in ABCWY (0, 2 month schedule) is measured in terms of number of participants achieving a 4-fold rise in hSBA titers against serogroups A, C, W and Y. The 4-fold rise is defined as: -a post-vaccination hSBA titer ≥ 16 for participants with a pre-vaccination hSBA titer < 4, -a post-vaccination hSBA titer ≥ 4 times the lower limit of quantitation (LLOQ) for participants with a pre-vaccination hSBA titer ≥LOD but <LLOQ, and. -a post-vaccination hSBA titer ≥ 4 times the pre-vaccination hSBA titer for participants with a pre-vaccination hSBA titer ≥LLOQ.
Time Frame: At Day 211 for ABCWY groups (1 month after the last MenABCWY-2Gen vaccination) and at Day 31 for Control group (1 month after the last MenACWY vaccination)
Population: Analysis was performed on the Phase II FSF, Per Protocol Set (PPS), which included all participants who received at least one dose of the study treatment to which they are randomised and have post-vaccination data (Full Analysis Set) for the specified analysis at specified timepoints minus participants with protocol deviations that lead to exclusion from the Per Protocol Set.
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_06 Group | ABCWY High dose_02 Group | Control Group
Number analyzed (Participants) | 135 | 116 | 147 | 118 | 159
Participants
  Men A: number analyzed (Participants) | 132 | 109 | 140 | 112 | 156
  Men A | 125 | 105 | 136 | 107 | 143
  Men C: number analyzed (Participants) | 135 | 113 | 146 | 118 | 152
  Men C | 129 | 107 | 132 | 111 | 92
  Men W: number analyzed (Participants) | 134 | 114 | 143 | 116 | 156
  Men W | 129 | 108 | 135 | 105 | 102
  Men Y: number analyzed (Participants) | 131 | 116 | 147 | 115 | 159
  Men Y | 122 | 102 | 131 | 100 | 95
Statistical Analysis 1: Comparison: ABCWY Low dose_06 Group vs Control Group; To demonstrate the immunological non-inferiority of the MenABCWY-2Gen vaccine (low dose) administered at 0,6-months schedule compared to the MenACWY vaccine administered at month 0 in the control group (Men A); Test type: Non-Inferiority — Non-inferiority (NI) was to be demonstrated if the lower limit of the 2-sided 97.5% CI for the difference in percentages of participants achieving a 4-fold rise in hSBA titres is above -10% at 1 month after the last MenABCWY-2Gen vaccination in the ABCWY low dose_06 group compared to the MenACWY vaccination in the Control group; Difference in percentage = 3.03, 97.5% CI 2-sided [-4.21 to 10.17] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: ABCWY Low dose_02 Group vs Control Group; To demonstrate the immunological non-inferiority of the MenABCWY-2Gen vaccine (low dose) administered at 0,2-months schedule compared to the MenACWY vaccine administered at month 0 in the control group (Men A); Test type: Non-Inferiority — NI was to be demonstrated if the lower limit of the 2-sided 97.5% CI for the difference in percentages of participants achieving a 4-fold rise in hSBA titres is above -10% at 1 month after the last MenABCWY-2Gen vaccination in the ABCWY low dose_02 group compared to the MenACWY vaccination in the Control group; Difference in percentage = 4.66, 97.5% CI 2-sided [-2.71 to 11.64] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 3: Comparison: ABCWY High dose_06 Group vs Control Group; To demonstrate the immunological non-inferiority of the MenABCWY-2Gen vaccine (high dose) administered at 0,6-months schedule compared to the MenACWY vaccine administered at month 0 in the control group (Men A); Test type: Non-Inferiority — NI was to be demonstrated if the lower limit of the 2-sided 97.5% CI for the difference in percentages of participants achieving a 4-fold rise in hSBA titres is above -10% at 1 month after the last MenABCWY-2Gen vaccination in the ABCWY high dose_06 group compared to the MenACWY vaccination in the Control group; Difference in percentage = 5.48, 97.5% CI 2-sided [-0.71 to 12.25] — [estimate comment as in outcome 10, analysis 3]
Statistical Analysis 4: Comparison: ABCWY High dose_02 Group vs Control Group; To demonstrate the immunological non-inferiority of the MenABCWY-2Gen vaccine (high dose) administered at 0,2-months schedule compared to the MenACWY vaccine administered at month 0 in the control group (Men A); Test type: Non-Inferiority — NI was to be demonstrated if the lower limit of the 2-sided 97.5% CI for the difference in percentages of participants achieving a 4-fold rise in hSBA titres is above -10% at 1 month after the last MenABCWY-2Gen vaccination in the ABCWY high dose_02 group compared to the MenACWY vaccination in the Control group; Difference in percentage = 3.87, 97.5% CI 2-sided [-3.70 to 10.97] — [estimate comment as in outcome 10, analysis 4]
Statistical Analysis 5: Comparison: ABCWY Low dose_06 Group vs Control Group; To demonstrate the immunological non-inferiority of the MenABCWY-2Gen vaccine (low dose) administered at 0,6-months schedule compared to the MenACWY vaccine administered at month 0 in the control group (Men C); Test type: Non-Inferiority — [test comment as in outcome 11, analysis 1]; Difference in percentage = 35.03, 97.5% CI 2-sided [25.22 to 44.75] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 6: Comparison: ABCWY Low dose_02 Group vs Control Group; To demonstrate the immunological non-inferiority of the MenABCWY-2Gen vaccine (low dose) administered at 0,2-months schedule compared to the MenACWY vaccine administered at month 0 in the control group (Men C); Test type: Non-Inferiority — [test comment as in outcome 11, analysis 2]; Difference in percentage = 34.16, 97.5% CI 2-sided [23.76 to 44.10] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 7: Comparison: ABCWY High dose_06 Group vs Control Group; To demonstrate the immunological non-inferiority of the MenABCWY-2Gen vaccine (high dose) administered at 0,6-months schedule compared to the MenACWY vaccine administered at month 0 in the control group (Men C); Test type: Non-Inferiority — [test comment as in outcome 11, analysis 3]; Difference in percentage = 29.88, 97.5% CI 2-sided [19.26 to 40.19] — [estimate comment as in outcome 10, analysis 3]
Statistical Analysis 8: Comparison: ABCWY High dose_02 Group vs Control Group; To demonstrate the immunological non-inferiority of the MenABCWY-2Gen vaccine (high dose) administered at 0,2-months schedule compared to the MenACWY vaccine administered at month 0 in the control group (Men C); Test type: Non-Inferiority — [test comment as in outcome 11, analysis 4]; Difference in percentage = 33.54, 97.5% CI 2-sided [23.09 to 43.54] — [estimate comment as in outcome 10, analysis 4]
Statistical Analysis 9: Comparison: ABCWY Low dose_06 Group vs Control Group; To demonstrate the immunological non-inferiority of the MenABCWY-2Gen vaccine (low dose) administered at 0,6-months schedule compared to the MenACWY vaccine administered at month 0 in the control group (Men W); Test type: Non-Inferiority — [test comment as in outcome 11, analysis 1]; Difference in percentage = 30.88, 97.5% CI 2-sided [21.61 to 40.32] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 10: Comparison: ABCWY Low dose_02 Group vs Control Group; To demonstrate the immunological non-inferiority of the MenABCWY-2Gen vaccine (low dose) administered at 0,2-months schedule compared to the MenACWY vaccine administered at month 0 in the control group (Men W); Test type: Non-Inferiority — NI was to be demonstrated if the lower limit of the 2-sided 97.5% CI for the difference in percentages of participants achieving a 4-fold rise in hSBA titres is above -10% at 1 month after the MenABCWY-2Gen MenACWY vaccination in the ABCWY low dose_02 group compared to the MenACWY vaccination in the Control group; Difference in percentage = 29.35, 97.5% CI 2-sided [19.31 to 39.08] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 11: Comparison: ABCWY High dose_06 Group vs Control Group; To demonstrate the immunological non-inferiority of the MenABCWY-2Gen vaccine (high dose) administered at 0,6-months schedule compared to the MenACWY vaccine administered at month 0 in the control group (Men W); Test type: Non-Inferiority — [test comment as in outcome 11, analysis 3]; Difference in percentage = 29.02, 97.5% CI 2-sided [19.42 to 38.67] — [estimate comment as in outcome 10, analysis 3]
Statistical Analysis 12: Comparison: ABCWY High dose_02 Group vs Control Group; To demonstrate the immunological non-inferiority of the MenABCWY-2Gen vaccine (high dose) administered at 0,2-months schedule compared to the MenACWY vaccine administered at month 0 in the control group (Men W); Test type: Non-Inferiority — [test comment as in outcome 11, analysis 4]; Difference in percentage = 25.13, 97.5% CI 2-sided [14.20 to 35.45] — [estimate comment as in outcome 10, analysis 4]
Statistical Analysis 13: Comparison: ABCWY Low dose_06 Group vs Control Group; To demonstrate the immunological non-inferiority of the MenABCWY-2Gen vaccine (low dose) administered at 0,6-months schedule compared to the MenACWY vaccine administered at month 0 in the control group (Men Y); Test type: Non-Inferiority — [test comment as in outcome 11, analysis 1]; Difference in percentage = 33.38, 97.5% CI 2-sided [23.08 to 43.26] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 14: Comparison: ABCWY Low dose_02 Group vs Control Group; To demonstrate the immunological non-inferiority of the MenABCWY-2Gen vaccine (low dose) administered at 0,2-months schedule compared to the MenACWY vaccine administered at month 0 in the control group (Men Y); Test type: Non-Inferiority — [test comment as in outcome 11, analysis 2]; Difference in percentage = 28.18, 97.5% CI 2-sided [16.61 to 38.86] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 15: Comparison: ABCWY High dose_06 Group vs Control Group; To demonstrate the immunological non-inferiority of the MenABCWY-2Gen vaccine (high dose) administered at 0,6-months schedule compared to the MenACWY vaccine administered at month 0 in the control group (Men Y); Test type: Non-Inferiority — [test comment as in outcome 11, analysis 3]; Difference in percentage = 29.37, 97.5% CI 2-sided [18.67 to 39.63] — [estimate comment as in outcome 10, analysis 3]
Statistical Analysis 16: Comparison: ABCWY High dose_02 Group vs Control Group; To demonstrate the immunological non-inferiority of the MenABCWY-2Gen vaccine (high dose) administered at 0,2-months schedule compared to the MenACWY vaccine administered at month 0 in the control group (Men Y); Test type: Non-Inferiority — [test comment as in outcome 11, analysis 4]; Difference in percentage = 27.21, 97.5% CI 2-sided [15.46 to 38.02] — [estimate comment as in outcome 10, analysis 4]

12. Primary Outcome: Number of Participants With Solicited Administration Site Events in Study Phase II (Formulation and Schedule-finding)
Description: Assessed solicited administration site events included injection site pain, erythema (redness), swelling and induration. Any = occurrence of the event regardless of intensity grade.
Time Frame: During the 7 days (including the day of vaccination) following vaccination at Day 1
Population: Analysis was performed on the Phase II FSF, Exposed set, which included all participants who received at least one dose of the study treatment and have post-vaccination data for the specified analysis at specified timepoints. Allocation per group using the enrolled set is based on the treatment administered.
Measure: Count of Participants; unit: Participants
Groups:
- Control (MenACWY) Group: Participants randomized to Control Group received a single dose of Menveo (MenACWY) on Day 1 during study Phase II (Formulation and Schedule-finding).
- Control (MenB_06) Group: Participants randomized to Control Group received 2 doses of Bexsero (MenB) vaccine on Day 1 and Day 181 following in a 0, 6- month schedule during study Phase II (Formulation and Schedule-finding).
Arm/Group | ABCWY Low dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_06 Group | ABCWY High dose_02 Group | Control (MenACWY) Group | Control (MenB_06) Group
Number analyzed (Participants) | 239 | 181 | 238 | 194 | 178 | 178
Participants
  Erythema | 32 | 0 | 29 | 0 | 6 | 13
  Induration | 22 | 1 | 30 | 1 | 6 | 11
  Pain | 217 | 39 | 220 | 42 | 76 | 145
  Swelling | 34 | 0 | 32 | 0 | 4 | 8

13. Primary Outcome: Number of Participants With Solicited Administration Site Events in Study Phase II (Formulation and Schedule-finding)
Description: as for outcome 12
Time Frame: During the 7 days (including the day of vaccination) following vaccination at Day 121
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_06 Group | ABCWY High dose_02 Group | Control (MenACWY) Group | Control (MenB_06) Group
Number analyzed (Participants) | 220 | 170 | 224 | 182 | 0 | 0
Participants
  Erythema (mm) | 0 | 17 | 0 | 14 |  |
  Induration (mm) | 1 | 15 | 0 | 18 |  |
  Pain | 28 | 143 | 26 | 153 |  |
  Swelling (mm) | 1 | 21 | 0 | 21 |  |

14. Primary Outcome: Number of Participants With Solicited Administration Site Events in Study Phase II (Formulation and Schedule-finding)
Description: as for outcome 12
Time Frame: During the 7 days (including the day of vaccination) following vaccination at Day 181
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_06 Group | ABCWY High dose_02 Group | Control (MenACWY) Group | Control (MenB_06) Group
Number analyzed (Participants) | 216 | 163 | 220 | 176 | 0 | 187
Participants
  Erythema | 23 | 15 | 21 | 17 |  | 18
  Induration | 18 | 17 | 20 | 15 |  | 16
  Pain | 191 | 134 | 187 | 146 |  | 154
  Swelling | 27 | 25 | 27 | 23 |  | 23

15. Primary Outcome: Number of Participants With Solicited Systemic Events in Study Phase II (Formulation and Schedule-finding)
Description: Assessed solicited systemic events included fever (temperature ≥ 38.0°C), nausea, fatigue, myalgia, arthralgia and headache. Any = occurrence of the event regardless of intensity grade or relation to the study vaccination.
Time Frame: During the 7 days (including the day of vaccination) following vaccination at Day 1
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_06 Group | ABCWY High dose_02 Group | Control Group
Number analyzed (Participants) | 239 | 181 | 238 | 194 | 197
Participants
  Arthralgia | 17 | 6 | 16 | 6 | 11
  Fatigue | 123 | 60 | 109 | 73 | 91
  Headache | 92 | 60 | 102 | 63 | 78
  Myalgia | 28 | 6 | 23 | 9 | 18
  Nausea | 30 | 16 | 23 | 13 | 19
  Fever (C) | 4 | 2 | 8 | 1 | 8

16. Primary Outcome: Number of Participants With Solicited Systemic Events in Study Phase II (Formulation and Schedule-finding)
Description: as for outcome 15
Time Frame: During the 7 days (including the day of vaccination) following vaccination at Day 121
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_06 Group | ABCWY High dose_02 Group | Control Group
Number analyzed (Participants) | 220 | 170 | 224 | 182 | 0
Participants
  Arthralgia | 2 | 13 | 4 | 8 |
  Fatigue | 46 | 72 | 42 | 68 |
  Headache | 46 | 56 | 47 | 58 |
  Myalgia | 4 | 21 | 8 | 23 |
  Nausea | 13 | 8 | 14 | 19 |
  Fever (C) | 1 | 5 | 2 | 5 |

17. Primary Outcome: Number of Participants With Solicited Systemic Events in Study Phase II (Formulation and Schedule-finding)
Description: as for outcome 15
Time Frame: During the 7 days (including the day of vaccination) following vaccination at Day 181
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_06 Group | ABCWY High dose_02 Group | Control Group
Number analyzed (Participants) | 216 | 163 | 220 | 176 | 187
Participants
  Arthralgia | 14 | 8 | 22 | 13 | 6
  Fatigue | 86 | 59 | 98 | 62 | 75
  Headache | 75 | 59 | 90 | 59 | 64
  Myalgia | 26 | 18 | 36 | 20 | 33
  Nausea | 22 | 11 | 31 | 12 | 15
  Fever (C) | 4 | 6 | 8 | 3 | 5

18. Primary Outcome: Number of Participants With Any Unsolicited AEs (Including All SAEs, AEs Leading to Withdrawal, and AESIs) in Study Phase II (Formulation and Schedule-finding)
Description: as for outcome 5
Time Frame: During the 30 days (including the day of vaccination) following vaccination at Day 1
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_06 Group | ABCWY High dose_02 Group | Control Group
Number analyzed (Participants) | 239 | 181 | 238 | 194 | 197
Participants | 51 | 34 | 52 | 35 | 27

19. Primary Outcome: Number of Participants With Any Unsolicited AEs (Including All SAEs, AEs Leading to Withdrawal, and AESIs) in Study Phase II (Formulation and Schedule-finding)
Description: as for outcome 5
Time Frame: During the 30 days (including the day of vaccination) following vaccination at Day 121
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_06 Group | ABCWY High dose_02 Group | Control Group
Number analyzed (Participants) | 220 | 170 | 224 | 182 | 0
Participants | 16 | 19 | 22 | 18 |

20. Primary Outcome: Number of Participants With Any Unsolicited AEs (Including All SAEs, AEs Leading to Withdrawal, and AESIs) in Study Phase II (Formulation and Schedule-finding)
Description: as for outcome 5
Time Frame: During the 30 days (including the day of vaccination) following vaccination at Day 181
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_06 Group | ABCWY High dose_02 Group | Control Group
Number analyzed (Participants) | 216 | 163 | 220 | 176 | 187
Participants | 28 | 24 | 42 | 27 | 28

21. Primary Outcome: Number of Participants With SAEs, AEs Leading to Withdrawal and AESIs in Study Phase II (Formulation and Schedule-Finding)
Description: as for outcome 7
Time Frame: Throughout the Phase II FSF study period (Day 1 through Day 541)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_06 Group | ABCWY High dose_02 Group | Control Group
Number analyzed (Participants) | 239 | 181 | 238 | 194 | 197
Participants
  SAEs | 9 | 7 | 4 | 4 | 2
  AEs leading to withdrawal | 1 | 0 | 1 | 1 | 0
  AESIs | 4 | 1 | 2 | 0 | 1

22. Primary Outcome: Number of Participants With Solicited Administration Site Events in Study Phase II (Sourcing)
Description: as for outcome 12
Time Frame: During the 7 days (including the day of vaccination) following vaccination at Day 1
Population: Analysis was performed on the Phase II Sourcing, Exposed set, which included all participants who received at least one dose of the study treatment and have post-vaccination data for the specified analysis at specified timepoints. Allocation per group using the enrolled set is based on the treatment administered.
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low dose_01 Group | ABCWY High dose_01 Group | ABCWY Low doseS_02 Group | ABCWY High doseS_02 Group | ABCWY Low doseS_06 Group | ABCWY High doseS_06 Group
Number analyzed (Participants) | 54 | 53 | 62 | 62 | 62 | 63
Participants
  Erythema | 0 | 0 | 0 | 0 | 0 | 0
  Induration | 0 | 0 | 0 | 0 | 0 | 0
  Pain | 2 | 4 | 3 | 1 | 1 | 2
  Swelling | 0 | 0 | 0 | 0 | 0 | 0

23. Primary Outcome: Number of Participants With Solicited Administration Site Events in Study Phase II (Sourcing)
Description: as for outcome 12
Time Frame: During the 7 days (including the day of vaccination) following vaccination at Day 31
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low dose_01 Group | ABCWY High dose_01 Group
Number analyzed (Participants) | 50 | 47
Participants
  Erythema | 0 | 1
  Induration | 0 | 0
  Pain | 0 | 1
  Swelling | 0 | 1

24. Primary Outcome: Number of Participants With Solicited Administration Site Events in Study Phase II (Sourcing)
Description: as for outcome 12
Time Frame: During the 7 days (including the day of vaccination) following vaccination at Day 61
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low doseS_02 Group | ABCWY High doseS_02 Group
Number analyzed (Participants) | 58 | 60
Participants
  Erythema | 0 | 0
  Induration | 0 | 0
  Pain | 2 | 3
  Swelling | 0 | 0

25. Primary Outcome: Number of Participants With Solicited Administration Site Events in Study Phase II (Sourcing)
Description: as for outcome 12
Time Frame: During the 7 days (including the day of vaccination) following vaccination at Day 181
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low doseS_06 Group | ABCWY High doseS_06 Group
Number analyzed (Participants) | 60 | 55
Participants
  Erythema | 0 | 0
  Induration | 0 | 0
  Pain | 4 | 3
  Swelling | 0 | 0

26. Primary Outcome: Number of Participants With Solicited Systemic Events in Study Phase II (Sourcing)
Description: as for outcome 15
Time Frame: During the 7 days (including the day of vaccination) following vaccination at Day 1
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low dose_01 Group | ABCWY High dose_01 Group | ABCWY Low doseS_02 Group | ABCWY High doseS_02 Group | ABCWY Low doseS_06 Group | ABCWY High doseS_06 Group
Number analyzed (Participants) | 54 | 53 | 62 | 62 | 62 | 63
Participants
  Arthralgia | 1 | 0 | 1 | 0 | 0 | 0
  Fatigue | 2 | 1 | 2 | 0 | 0 | 1
  Headache | 3 | 0 | 0 | 0 | 0 | 3
  Myalgia | 1 | 0 | 1 | 0 | 0 | 1
  Nausea | 2 | 1 | 0 | 0 | 1 | 0
  Fever (C) | 0 | 0 | 0 | 0 | 0 | 0

27. Primary Outcome: Number of Participants With Solicited Systemic Events in Study Phase II (Sourcing)
Description: as for outcome 15
Time Frame: During the 7 days (including the day of vaccination) following vaccination at Day 31
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low dose_01 Group | ABCWY High dose_01 Group
Number analyzed (Participants) | 50 | 47
Participants
  Arthralgia | 0 | 0
  Fatigue | 1 | 0
  Headache | 0 | 3
  Myalgia | 0 | 0
  Nausea | 0 | 2
  Fever (C) | 0 | 0

28. Primary Outcome: Number of Participants With Solicited Systemic Events in Study Phase II (Sourcing)
Description: as for outcome 15
Time Frame: During the 7 days (including the day of vaccination) following vaccination at Day 61
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low doseS_02 Group | ABCWY High doseS_02 Group
Number analyzed (Participants) | 58 | 60
Participants
  Arthralgia | 0 | 0
  Fatigue | 0 | 0
  Headache | 0 | 0
  Myalgia | 1 | 0
  Nausea | 0 | 0
  Fever (C) | 0 | 0

29. Primary Outcome: Number of Participants With Solicited Systemic Events in Study Phase II (Sourcing)
Description: as for outcome 15
Time Frame: During the 7 days (including the day of vaccination) following vaccination at Day 181
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low doseS_06 Group | ABCWY High doseS_06 Group
Number analyzed (Participants) | 60 | 55
Participants
  Arthralgia | 0 | 0
  Fatigue | 0 | 0
  Headache | 0 | 0
  Myalgia | 0 | 0
  Nausea | 0 | 0
  Fever (C) | 0 | 0

30. Primary Outcome: Number of Participants With Any Unsolicited AEs (Including All SAEs, AEs Leading to Withdrawal, and AESIs) in Study Phase II (Sourcing)
Description: as for outcome 5
Time Frame: During the 30 days (including the day of vaccination) following vaccination at Day 1
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low dose_01 Group | ABCWY High dose_01 Group | ABCWY Low doseS_02 Group | ABCWY High doseS_02 Group | ABCWY Low doseS_06 Group | ABCWY High doseS_06 Group
Number analyzed (Participants) | 54 | 53 | 62 | 62 | 62 | 63
Participants | 10 | 12 | 14 | 8 | 10 | 18

31. Primary Outcome: Number of Participants With Any Unsolicited AEs (Including All SAEs, AEs Leading to Withdrawal, and AESIs) in Study Phase II (Sourcing)
Description: as for outcome 5
Time Frame: During the 30 days (including the day of vaccination) following vaccination at Day 31
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low dose_01 Group | ABCWY High dose_01 Group
Number analyzed (Participants) | 50 | 47
Participants | 11 | 16

32. Primary Outcome: Number of Participants With Any Unsolicited AEs (Including All SAEs, AEs Leading to Withdrawal, and AESIs) in Study Phase II (Sourcing)
Description: as for outcome 5
Time Frame: During the 30 days (including the day of vaccination) following vaccination at Day 61
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low doseS_02 Group | ABCWY High doseS_02 Group
Number analyzed (Participants) | 58 | 60
Participants | 8 | 7

33. Primary Outcome: Number of Participants With Any Unsolicited AEs (Including All SAEs, AEs Leading to Withdrawal, and AESIs) in Study Phase II (Sourcing)
Description: as for outcome 5
Time Frame: During the 30 days (including the day of vaccination) following vaccination at Day 181
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low doseS_06 Group | ABCWY High doseS_06 Group
Number analyzed (Participants) | 60 | 55
Participants | 10 | 9

34. Primary Outcome: Number of Participants With SAEs, AEs Leading to Withdrawal and AESIs in Study Phase II (Sourcing)
Description: as for outcome 7
Time Frame: Throughout the study period (Day 1 through Day 211)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low dose_01 Group | ABCWY High dose_01 Group
Number analyzed (Participants) | 54 | 53
Participants
  SAEs | 0 | 0
  AEs leading to withdrawal | 0 | 0
  AESIs | 0 | 0

35. Primary Outcome: Number of Participants With SAEs, AEs Leading to Withdrawal and AESIs in Study Phase II (Sourcing)
Description: as for outcome 7
Time Frame: Throughout the study period (Day 1 through Day 241)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low doseS_02 Group | ABCWY High doseS_02 Group
Number analyzed (Participants) | 62 | 62
Participants
  SAEs | 2 | 1
  AEs leading to withdrawal | 1 | 0
  AESIs | 0 | 1

36. Primary Outcome: Number of Participants With SAEs, AEs Leading to Withdrawal and AESIs in Study Phase II (Sourcing)
Description: as for outcome 7
Time Frame: Throughout the study period (Day 1 through Day 361)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low doseS_06 Group | ABCWY High doseS_06 Group
Number analyzed (Participants) | 62 | 63
Participants
  SAEs | 0 | 4
  AEs leading to withdrawal | 0 | 2
  AESIs | 0 | 0

37. Secondary Outcome: Percentage of Participants Classified by Percentages of Serogroup B Invasive Disease Strains Killed Using Enc-hSBA in Each Participant in Study Phase II (Formulation and Schedule-finding)
Description: The percentages of strains killed measured by enc-hSBA against a randomly selected panel of strains and the corresponding exact 2-sided 95% CIs based on Clopper-Pearson method is calculated in all groups at 1 month after the last vaccination of MenABCWY-2Gen (low and high dose) vaccine administered at 0,2 and 0,6-months schedule and of the MenB vaccine administered at 0,6-months schedule.
Time Frame: At Day 211 (1 month after the last vaccination)
Population: Analysis was performed on the Phase II FSF Full Analysis Set, which included all participants at least 1 dose of the study intervention and have post-vaccination immunogenicity data for the specified analysis at specified timepoints. The allocation in a group is done in function of the randomised intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ABCWY Low dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_06 Group | ABCWY High dose_02 Group | Control Group
Number analyzed (Participants) | 205 | 161 | 215 | 169 | 176
Percentage of participants
  >= (greater than/equal to) 50% killed strains | 98.5 [95.8 to 99.7] | 97.5 [93.8 to 99.3] | 97.7 [94.7 to 99.2] | 98.8 [95.8 to 99.9] | 98.3 [95.1 to 99.6]
  >=55% killed strains | 98.0 [95.1 to 99.5] | 95.7 [91.2 to 98.2] | 97.7 [94.7 to 99.2] | 98.2 [94.9 to 99.6] | 96.6 [92.7 to 98.7]
  >=60% killed strains | 96.6 [93.1 to 98.6] | 95.0 [90.4 to 97.8] | 97.2 [94.0 to 99.0] | 97.0 [93.2 to 99.0] | 95.5 [91.2 to 98.0]
  >=65% killed strains | 95.6 [91.8 to 98.0] | 92.5 [87.3 to 96.1] | 96.3 [92.8 to 98.4] | 95.9 [91.7 to 98.3] | 93.8 [89.1 to 96.8]
  >=70% killed strains | 94.1 [90.0 to 96.9] | 89.4 [83.6 to 93.7] | 94.4 [90.5 to 97.1] | 94.7 [90.1 to 97.5] | 88.6 [83.0 to 92.9]
  >=75% killed strains | 91.2 [86.5 to 94.7] | 82.0 [75.2 to 87.6] | 90.2 [85.5 to 93.9] | 88.8 [83.0 to 93.1] | 80.7 [74.1 to 86.2]
  >=80% killed strains | 88.8 [83.6 to 92.8] | 77.6 [70.4 to 83.8] | 87.4 [82.3 to 91.6] | 82.8 [76.3 to 88.2] | 75.6 [68.5 to 81.7]
  >=85% killed strains | 82.9 [77.1 to 87.8] | 64.6 [56.7 to 72.0] | 82.8 [77.1 to 87.6] | 75.1 [67.9 to 81.5] | 63.6 [56.1 to 70.7]
  >=90% killed strains | 71.2 [64.5 to 77.3] | 53.4 [45.4 to 61.3] | 70.7 [64.1 to 76.7] | 55.0 [47.2 to 62.7] | 52.3 [44.6 to 59.8]
  >=95% killed strains | 43.4 [36.5 to 50.5] | 29.2 [22.3 to 36.9] | 44.2 [37.4 to 51.1] | 34.3 [27.2 to 42.0] | 26.1 [19.8 to 33.3]
  100% killed strains | 23.4 [17.8 to 29.8] | 14.3 [9.3 to 20.7] | 24.2 [18.6 to 30.5] | 17.2 [11.8 to 23.7] | 15.3 [10.4 to 21.5]

38. Secondary Outcome: Number of Participants With hSBA Titers ≥ LLOQ for Each and All Serogroup B Indicator Strains in Study Phase II (Formulation and Schedule-finding)
Description: The immune response to MenABCWY-2Gen (low and high dose) administered at 0,2 and 0,6-months schedule and MenB vaccine administered at 0,6-months schedule is evaluated by measuring bactericidal activity using a qualified AO hSBA against a standard panel of serogroup B indicator strains.
Time Frame: At Day 1 in ABCWY (0,6-months) and Control groups, Day 31 in ABCWY groups (0,2-months) and Day 211 in all study groups
Population: as for outcome 37
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low dose_06 Group | ABCWY High dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_02 Group | Control Group
Number analyzed (Participants) | 209 | 214 | 173 | 189 | 194
Participants
  fHbp, Day 1: number analyzed (Participants) | 209 | 214 | 0 | 0 | 194
  fHbp, Day 1 | 9 | 10 |  |  | 12
  fHbp, Day 31: number analyzed (Participants) | 0 | 0 | 173 | 189 | 0
  fHbp, Day 31 |  |  | 14 | 14 |
  fHbp, Day 211: number analyzed (Participants) | 201 | 213 | 159 | 168 | 179
  fHbp, Day 211 | 175 | 184 | 112 | 137 | 137
  NadA, Day 1: number analyzed (Participants) | 201 | 211 | 0 | 0 | 189
  NadA, Day 1 | 16 | 23 |  |  | 14
  NadA, Day 31: number analyzed (Participants) | 0 | 0 | 168 | 185 | 0
  NadA, Day 31 |  |  | 18 | 14 |
  NadA, Day 211: number analyzed (Participants) | 197 | 201 | 150 | 162 | 171
  NadA, Day 211 | 175 | 169 | 120 | 131 | 147
  NHBA, Day 1: number analyzed (Participants) | 207 | 213 | 0 | 0 | 189
  NHBA, Day 1 | 43 | 49 |  |  | 40
  NHBA, Day 31: number analyzed (Participants) | 0 | 0 | 172 | 186 | 0
  NHBA, Day 31 |  |  | 46 | 44 |
  NHBA, Day 211: number analyzed (Participants) | 199 | 212 | 155 | 167 | 177
  NHBA, Day 211 | 197 | 208 | 148 | 163 | 172
  PorA, Day 1: number analyzed (Participants) | 208 | 213 | 0 | 0 | 190
  PorA, Day 1 | 7 | 9 |  |  | 8
  PorA, Day 31: number analyzed (Participants) | 0 | 0 | 161 | 173 | 0
  PorA, Day 31 |  |  | 8 | 8 |
  PorA, Day 211: number analyzed (Participants) | 200 | 214 | 153 | 169 | 178
  PorA, Day 211 | 171 | 179 | 106 | 136 | 136
  fHbp V1.13, Day 1: number analyzed (Participants) | 203 | 209 | 0 | 0 | 184
  fHbp V1.13, Day 1 | 32 | 31 |  |  | 34
  fHbp V1.13, Day 31: number analyzed (Participants) | 0 | 0 | 171 | 184 | 0
  fHbp V1.13, Day 31 |  |  | 31 | 31 |
  fHbp V1.13, Day 211: number analyzed (Participants) | 188 | 194 | 142 | 148 | 168
  fHbp V1.13, Day 211 | 162 | 169 | 97 | 111 | 130
  fHbp V2, Day 1: number analyzed (Participants) | 203 | 209 | 0 | 0 | 185
  fHbp V2, Day 1 | 8 | 12 |  |  | 13
  fHbp V2, Day 31: number analyzed (Participants) | 0 | 0 | 171 | 184 | 0
  fHbp V2, Day 31 |  |  | 12 | 21 |
  fHbp V2, Day 211: number analyzed (Participants) | 195 | 204 | 150 | 161 | 172
  fHbp V2, Day 211 | 186 | 192 | 128 | 144 | 72
  fHbp V3, Day 1: number analyzed (Participants) | 203 | 209 | 0 | 0 | 185
  fHbp V3, Day 1 | 15 | 16 |  |  | 11
  fHbp V3, Day 31: number analyzed (Participants) | 0 | 0 | 172 | 184 | 0
  fHbp V3, Day 31 |  |  | 13 | 21 |
  fHbp V3, Day 211: number analyzed (Participants) | 194 | 204 | 151 | 162 | 172
  fHbp V3, Day 211 | 155 | 168 | 95 | 107 | 41
  Composite Response, Day 1: number analyzed (Participants) | 194 | 206 | 0 | 0 | 179
  Composite Response, Day 1 | 1 | 1 |  |  | 1
  Composite Response, Day 31: number analyzed (Participants) | 0 | 0 | 151 | 164 | 0
  Composite Response, Day 31 |  |  | 3 | 3 |
  Composite Response, Day 211: number analyzed (Participants) | 180 | 181 | 131 | 134 | 158
  Composite Response, Day 211 | 121 | 126 | 60 | 73 | 30

39. Secondary Outcome: Number of Participants With 4-fold Rise in hSBA Titers Against Serogroup B Indicator Strains in Study Phase II (Formulation and Schedule-finding)
Description: The immune response to MenABCWY-2Gen (low and high dose) vaccine when administered at 0,2- or 0,6-months schedule and to MenB vaccine administered at 0,6-months schedule, relative to day 1 in ABCWY (0,6 month schedule) and control groups and day 31 in ABCWY (0,2 month schedule) is measured in terms of number of participants achieving a 4-fold rise in hSBA titers against serogroup B indicator strains. The 4-fold rise is defined as: -a post-vaccination hSBA titer ≥ 16 for participants with a pre-vaccination hSBA titre < 4, -a post-vaccination hSBA titer ≥ 4 times the LLOQ for participants with a pre-vaccination hSBA titer ≥LOD but <LLOQ, and. -a post-vaccination hSBA titer ≥ 4 times the pre-vaccination hSBA titer for participants with a pre-vaccination hSBA titer ≥ LLOQ.
Time Frame: At Day 211 (1 month after the last vaccination)
Population: as for outcome 37
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_06 Group | ABCWY High dose_02 Group | Control Group
Number analyzed (Participants) | 178 | 155 | 193 | 168 | 177
Participants
  fHbp | 144 | 89 | 155 | 122 | 119
  NadA: number analyzed (Participants) | 166 | 141 | 179 | 159 | 167
  NadA | 135 | 104 | 133 | 113 | 135
  NHBA: number analyzed (Participants) | 174 | 150 | 191 | 164 | 171
  NHBA | 162 | 122 | 175 | 136 | 139
  PorA: number analyzed (Participants) | 175 | 140 | 193 | 157 | 172
  PorA | 124 | 69 | 133 | 92 | 109
  fHbp V1.13: number analyzed (Participants) | 162 | 137 | 173 | 144 | 158
  fHbp V1.13 | 126 | 82 | 140 | 92 | 97
  fHbp V2: number analyzed (Participants) | 168 | 144 | 182 | 157 | 163
  fHbp V2 | 119 | 69 | 138 | 91 | 21
  fHbp V3: number analyzed (Participants) | 167 | 146 | 182 | 158 | 163
  fHbp V3 | 92 | 62 | 120 | 77 | 7

40. Secondary Outcome: hSBA Geometric Mean Titers (GMTs) Against Serogroup B Indicator Strains in Study Phase II (Formulation and Schedule-finding)
Description: For each B strains, the GMTs are calculated with their associated 2-sided 95% CIs, by exponentiating the corresponding log-transformed means and their 95% CIs.
Time Frame: At Day 1 in ABCWY groups (0,6-months) and Control groups, Day 31 in ABCWY groups (0,2-months) and Day 211 in all study groups
Population: as for outcome 37
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ABCWY Low dose_06 Group | ABCWY High dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_02 Group | Control Group
Number analyzed (Participants) | 209 | 214 | 173 | 189 | 194
Titers
  fHbp, Day 1: number analyzed (Participants) | 209 | 214 | 0 | 0 | 194
  fHbp, Day 1 | 8.7 [8.1 to 9.3] | 8.8 [8.2 to 9.4] |  |  | 8.9 [8.3 to 9.6]
  fHbp, Day 31: number analyzed (Participants) | 0 | 0 | 173 | 189 | 0
  fHbp, Day 31 |  |  | 9.4 [8.7 to 10.1] | 9.5 [8.8 to 10.2] |
  fHbp, Day 211: number analyzed (Participants) | 201 | 213 | 159 | 168 | 179
  fHbp, Day 211 | 109.1 [86.0 to 138.3] | 140.2 [110.9 to 177.4] | 47.7 [37.0 to 61.5] | 82.4 [63.8 to 106.4] | 62.0 [48.3 to 79.5]
  NadA, Day 1: number analyzed (Participants) | 201 | 211 | 0 | 0 | 189
  NadA, Day 1 | 7.8 [7.2 to 8.4] | 8.1 [7.5 to 8.7] |  |  | 7.7 [7.1 to 8.3]
  NadA, Day 31: number analyzed (Participants) | 0 | 0 | 168 | 185 | 0
  NadA, Day 31 |  |  | 8.2 [7.6 to 8.9] | 8.1 [7.5 to 8.8] |
  NadA, Day 211: number analyzed (Participants) | 197 | 201 | 150 | 162 | 171
  NadA, Day 211 | 82.5 [64.8 to 105.1] | 88.5 [69.5 to 112.7] | 58.9 [45.2 to 76.7] | 56.8 [43.7 to 73.8] | 109.1 [84.5 to 140.9]
  NHBA, Day 1: number analyzed (Participants) | 207 | 213 | 0 | 0 | 189
  NHBA, Day 1 | 5.0 [4.2 to 6.0] | 5.2 [4.4 to 6.2] |  |  | 5.3 [4.4 to 6.4]
  NHBA, Day 31: number analyzed (Participants) | 0 | 0 | 172 | 186 | 0
  NHBA, Day 31 |  |  | 6.3 [5.3 to 7.7] | 6.0 [5.0 to 7.2] |
  NHBA, Day 211: number analyzed (Participants) | 199 | 212 | 155 | 167 | 177
  NHBA, Day 211 | 128.4 [106.4 to 155.0] | 169.5 [141.0 to 203.9] | 75.1 [61.4 to 91.9] | 101.0 [82.6 to 123.4] | 58.2 [47.9 to 70.7]
  PorA, Day 1: number analyzed (Participants) | 208 | 213 | 0 | 0 | 190
  PorA, Day 1 | 4.5 [4.2 to 4.8] | 4.4 [4.1 to 4.8] |  |  | 4.3 [4.0 to 4.6]
  PorA, Day 31: number analyzed (Participants) | 0 | 0 | 161 | 173 | 0
  PorA, Day 31 |  |  | 4.6 [4.3 to 5.0] | 4.6 [4.3 to 5.0] |
  PorA, Day 211: number analyzed (Participants) | 200 | 214 | 153 | 169 | 178
  PorA, Day 211 | 35.7 [28.3 to 45.2] | 41.1 [32.7 to 51.6] | 18.4 [14.3 to 23.7] | 28.2 [21.9 to 36.1] | 30.4 [23.9 to 38.8]
  fHbp V1.13, Day 1: number analyzed (Participants) | 203 | 209 | 0 | 0 | 184
  fHbp V1.13, Day 1 | 5.1 [4.3 to 6.1] | 5.2 [4.3 to 6.2] |  |  | 5.2 [4.3 to 6.3]
  fHbp V1.13, Day 31: number analyzed (Participants) | 0 | 0 | 171 | 184 | 0
  fHbp V1.13, Day 31 |  |  | 5.6 [4.6 to 6.7] | 5.8 [4.8 to 7.0] |
  fHbp V1.13, Day 211: number analyzed (Participants) | 188 | 194 | 142 | 148 | 168
  fHbp V1.13, Day 211 | 88.3 [63.4 to 122.9] | 122.1 [88.3 to 169.0] | 39.7 [27.8 to 56.7] | 54.9 [38.2 to 78.9] | 36.9 [26.3 to 51.9]
  fHbp V2, Day 1: number analyzed (Participants) | 203 | 209 | 0 | 0 | 185
  fHbp V2, Day 1 | 2.7 [2.5 to 2.9] | 2.7 [2.6 to 2.9] |  |  | 2.7 [2.6 to 2.9]
  fHbp V2, Day 31: number analyzed (Participants) | 0 | 0 | 171 | 184 | 0
  fHbp V2, Day 31 |  |  | 2.8 [2.7 to 3.0] | 3.0 [2.8 to 3.2] |
  fHbp V2, Day 211: number analyzed (Participants) | 195 | 204 | 150 | 161 | 172
  fHbp V2, Day 211 | 31.7 [25.2 to 39.8] | 44.0 [35.1 to 55.2] | 17.3 [13.5 to 22.1] | 23.2 [18.1 to 29.7] | 5.2 [4.1 to 6.6]
  fHbp V3, Day 1: number analyzed (Participants) | 203 | 209 | 0 | 0 | 185
  fHbp V3, Day 1 | 8.7 [7.9 to 9.5] | 8.7 [7.9 to 9.5] |  |  | 8.3 [7.5 to 9.1]
  fHbp V3, Day 31: number analyzed (Participants) | 0 | 0 | 172 | 184 | 0
  fHbp V3, Day 31 |  |  | 8.7 [7.9 to 9.6] | 8.9 [8.2 to 9.8] |
  fHbp V3, Day 211: number analyzed (Participants) | 194 | 204 | 151 | 162 | 172
  fHbp V3, Day 211 | 50.7 [40.4 to 63.7] | 65.7 [52.5 to 82.3] | 27.0 [21.1 to 34.4] | 33.2 [25.9 to 42.4] | 10.8 [8.6 to 13.7]

41. Secondary Outcome: hSBA Geometric Mean Ratios (GMRs) Against Serogroup B Indicator Strains in Study Phase II (Formulation and Schedule-finding)
Description: For each B strains, the GMRs (post-vaccination/ Baseline) are calculated with their associated 2-sided 95% CIs, by exponentiating the corresponding log-transformed means and their 95% CIs.
Time Frame: At Day 211 in all study groups versus Day 1 in ABCWY (0,6-months) and Control groups and Day 31 in ABCWY groups (0,2-months)
Population: as for outcome 37
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | ABCWY Low dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_06 Group | ABCWY High dose_02 Group | Control Group
Number analyzed (Participants) | 178 | 155 | 193 | 168 | 177
Ratio
  fHbp | 13.4 [10.5 to 17.2] | 5.6 [4.3 to 7.2] | 16.5 [12.9 to 21.0] | 9.0 [6.9 to 11.6] | 7.0 [5.5 to 9.1]
  NadA: number analyzed (Participants) | 166 | 141 | 179 | 159 | 167
  NadA | 11.1 [8.5 to 14.3] | 7.1 [5.4 to 9.3] | 10.8 [8.4 to 14.0] | 7.1 [5.4 to 9.3] | 14.7 [11.3 to 19.1]
  NHBA: number analyzed (Participants) | 174 | 150 | 191 | 164 | 171
  NHBA | 29.3 [23.5 to 36.7] | 14.0 [11.1 to 17.6] | 34.2 [27.5 to 42.5] | 18.4 [14.6 to 23.1] | 11.5 [9.1 to 14.4]
  PorA: number analyzed (Participants) | 175 | 140 | 193 | 157 | 172
  PorA | 8.6 [6.7 to 10.9] | 4.5 [3.5 to 5.8] | 10.1 [8.1 to 12.8] | 6.3 [4.9 to 8.1] | 7.4 [5.8 to 9.4]
  fHbp V1.13: number analyzed (Participants) | 162 | 137 | 173 | 144 | 158
  fHbp V1.13 | 17.8 [12.8 to 24.9] | 8.2 [5.8 to 11.7] | 24.9 [18.0 to 34.6] | 9.8 [6.9 to 14.0] | 7.0 [5.0 to 9.8]
  fHbp V2: number analyzed (Participants) | 168 | 144 | 182 | 157 | 163
  fHbp V2 | 12.7 [10.1 to 16.1] | 6.9 [5.4 to 8.8] | 17.1 [13.6 to 21.5] | 8.0 [6.2 to 10.2] | 2.0 [1.5 to 2.5]
  fHbp V3: number analyzed (Participants) | 167 | 146 | 182 | 158 | 163
  fHbp V3 | 5.9 [4.7 to 7.4] | 3.5 [2.7 to 4.4] | 7.7 [6.1 to 9.7] | 3.7 [2.9 to 4.8] | 1.3 [1.0 to 1.7]

42. Secondary Outcome: Number of Participants With hSBA Titers ≥ LLOQ for Serogroups A, C, W and Y in Study Phase II (Formulation and Schedule-finding)
Description: The number of participants with hSBA titers ≥ LLOQ and the corresponding exact 2-sided 95% CIs based on Clopper-Pearson method are calculated. Baseline (pre-vaccination) was evaluated at Day 1 for 0,6 schedules and Control, at Month 1 for 0,2 schedules. Post vaccination was evaluated at Month 7 for all MenABCWY groups, at Month 1 for Control group.
Time Frame: Day 1 in ABCWY (0,6 Months) & Control; Day 31 pre-vaccination in ABCWY (0,2 Months); Day 31 post-first MenABCWY-2Gen in ABCWY (0,6 Months); Day 211 post-last MenABCWY-2Gen in all ABCWY; Day 31 post-MenACWY in Control
Population: as for outcome 37
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low dose_06 Group | ABCWY High dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_02 Group | Control Group
Number analyzed (Participants) | 222 | 226 | 175 | 189 | 193
Participants
  Men A, Day 1: number analyzed (Participants) | 208 | 201 | 0 | 0 | 190
  Men A, Day 1 | 23 | 12 |  |  | 20
  Men A, Day 31 (Pre vaccination): number analyzed (Participants) | 0 | 0 | 170 | 184 | 0
  Men A, Day 31 (Pre vaccination) |  |  | 19 | 16 |
  Men A, Day 31 (Post vaccination): number analyzed (Participants) | 204 | 221 | 0 | 0 | 187
  Men A, Day 31 (Post vaccination) | 170 | 180 |  |  | 174
  Men A, Day 211 (Post vaccination): number analyzed (Participants) | 202 | 212 | 159 | 167 | 0
  Men A, Day 211 (Post vaccination) | 198 | 208 | 155 | 166 |
  Men C, Day 1: number analyzed (Participants) | 209 | 211 | 0 | 0 | 193
  Men C, Day 1 | 83 | 85 |  |  | 88
  Men C, Day 31 (Pre vaccination): number analyzed (Participants) | 0 | 0 | 173 | 189 | 0
  Men C, Day 31 (Pre vaccination) |  |  | 69 | 76 |
  Men C, Day 31 (Post vaccination): number analyzed (Participants) | 219 | 217 | 0 | 0 | 181
  Men C, Day 31 (Post vaccination) | 160 | 162 |  |  | 141
  Men C, Day 211 (Post vaccination): number analyzed (Participants) | 204 | 213 | 160 | 171 | 0
  Men C, Day 211 (Post vaccination) | 199 | 207 | 158 | 167 |
  Men W, Day 1: number analyzed (Participants) | 207 | 210 | 0 | 0 | 192
  Men W, Day 1 | 40 | 37 |  |  | 36
  Men W, Day 31 (Pre vaccination): number analyzed (Participants) | 0 | 0 | 173 | 187 | 0
  Men W, Day 31 (Pre vaccination) |  |  | 36 | 36 |
  Men W, Day 31 (Post vaccination): number analyzed (Participants) | 222 | 221 | 0 | 0 | 188
  Men W, Day 31 (Post vaccination) | 165 | 173 |  |  | 140
  Men W, Day 211 (Post vaccination): number analyzed (Participants) | 204 | 213 | 161 | 169 | 0
  Men W, Day 211 (Post vaccination) | 203 | 211 | 157 | 168 |
  Men Y, Day 1: number analyzed (Participants) | 207 | 211 | 0 | 0 | 193
  Men Y, Day 1 | 22 | 26 |  |  | 33
  Men Y, Day 31 (Pre vaccination): number analyzed (Participants) | 0 | 0 | 175 | 187 | 0
  Men Y, Day 31 (Pre vaccination) |  |  | 31 | 24 |
  Men Y, Day 31 (Post vaccination): number analyzed (Participants) | 222 | 226 | 0 | 0 | 190
  Men Y, Day 31 (Post vaccination) | 135 | 139 |  |  | 141
  Men Y, Day 211 (Post vaccination): number analyzed (Participants) | 203 | 214 | 161 | 169 | 0
  Men Y, Day 211 (Post vaccination) | 198 | 201 | 152 | 158 |

43. Secondary Outcome: Number of Participants With a 4-fold Rise in hSBA Titers Against Serogroups A, C, W and Y in Study Phase II (Formulation and Schedule-finding)
Description: The immune response to the MenABCWY-2Gen (low and high dose) vaccine when administered at 0,6-months schedule, relative to day 1 was measured in terms of percentage of participants achieving a 4-fold rise in hSBA titers against serogroups A, C, W and Y. Serum bactericidal activity against MenACWY were determined by using a validated AO hSBA. The 4-fold rise is defined as: -a post-vaccination hSBA titre ≥ 16 for participants with a pre-vaccination hSBA titre < 4, -a post-vaccination hSBA titre ≥ 4 times the LLOQ for participants with a pre-vaccination hSBA titre ≥ LOD but < LLOQ, and. -a post-vaccination hSBA titre ≥4 times the pre-vaccination hSBA titre for participants with a pre-vaccination hSBA titre ≥ LLOQ.
Time Frame: At Day 31 (1 month after the first MenABCWY-2Gen vaccination) in ABCWY (0,6-months) groups
Population: as for outcome 37
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Low dose_06 Group | ABCWY High dose_06 Group | Control Group
Number analyzed (Participants) | 194 | 201 | 186
Participants
  Men A: number analyzed (Participants) | 176 | 186 | 180
  Men A | 145 | 145 | 166
  Men C: number analyzed (Participants) | 193 | 192 | 178
  Men C | 125 | 119 | 113
  Men W: number analyzed (Participants) | 194 | 195 | 183
  Men W | 132 | 139 | 124
  Men Y: number analyzed (Participants) | 193 | 201 | 186
  Men Y | 105 | 104 | 116

44. Secondary Outcome: hSBA GMTs Against Serogroups A, C, W and Y in Study Phase II (Formulation and Schedule-finding)
Description: The immune response to the MenABCWY-2Gen (low and high dose) vaccine (0,2- and 0,6-months schedule) and MenACWY vaccine (single dose) was evaluated by hSBA titers which are logarithmically transformed (base10) to fulfil the normal distribution assumption. For each serogroup A, C, W and Y, the GMTs are calculated with their associated 2-sided 95% CIs, by exponentiating the corresponding log-transformed means and their 95% CIs.
Time Frame: as for outcome 42
Population: as for outcome 37
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ABCWY Low dose_06 Group | ABCWY High dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_02 Group | Control Group
Number analyzed (Participants) | 222 | 226 | 181 | 194 | 193
Titers
  Men A, Day 1: number analyzed (Participants) | 208 | 201 | 0 | 0 | 190
  Men A, Day 1 | 9.7 [8.5 to 11.2] | 8.7 [7.5 to 10.0] |  |  | 9.3 [8.0 to 10.7]
  Men A, Day 31 (Pre vaccination): number analyzed (Participants) | 0 | 0 | 181 | 194 | 0
  Men A, Day 31 (Pre vaccination) |  |  | 9.9 [8.5 to 11.4] | 8.7 [7.5 to 10.1] |
  Men A, Day 31 (Post vaccination): number analyzed (Participants) | 204 | 221 | 0 | 0 | 187
  Men A, Day 31 (Post vaccination) | 174.3 [127.6 to 238.1] | 169.5 [124.6 to 230.5] |  |  | 410.6 [299.0 to 564.1]
  Men A, Day 211 (Post vaccination): number analyzed (Participants) | 202 | 212 | 159 | 167 | 0
  Men A, Day 211 (Post vaccination) | 356.3 [296.7 to 427.9] | 422.8 [352.8 to 506.7] | 339.5 [278.9 to 413.1] | 356.9 [293.8 to 433.4] |
  Men C, Day 1: number analyzed (Participants) | 209 | 211 | 0 | 0 | 193
  Men C, Day 1 | 10.7 [8.6 to 13.3] | 10.3 [8.2 to 12.8] |  |  | 11.5 [9.2 to 14.3]
  Men C, Day 31 (Pre vaccination): number analyzed (Participants) | 0 | 0 | 173 | 189 | 0
  Men C, Day 31 (Pre vaccination) |  |  | 10.4 [8.3 to 13.1] | 10.9 [8.7 to 13.6] |
  Men C, Day 31 (Post vaccination): number analyzed (Participants) | 219 | 217 | 0 | 0 | 181
  Men C, Day 31 (Post vaccination) | 170.4 [106.8 to 272.0] | 162.0 [100.9 to 259.9] |  |  | 209.5 [128.4 to 341.9]
  Men C, Day 211 (Post vaccination): number analyzed (Participants) | 204 | 213 | 160 | 171 | 0
  Men C, Day 211 (Post vaccination) | 768.4 [601.2 to 982.0] | 738.9 [579.1 to 942.8] | 677.6 [521.0 to 881.2] | 652.5 [502.5 to 847.3] |
  Men W, Day 1: number analyzed (Participants) | 207 | 210 | 0 | 0 | 192
  Men W, Day 1 | 8.0 [6.5 to 9.9] | 7.2 [5.8 to 8.9] |  |  | 7.6 [6.1 to 9.5]
  Men W, Day 31 (Pre vaccination): number analyzed (Participants) | 0 | 0 | 173 | 187 | 0
  Men W, Day 31 (Pre vaccination) |  |  | 8.5 [6.8 to 10.7] | 8.1 [6.5 to 10.0] |
  Men W, Day 31 (Post vaccination): number analyzed (Participants) | 222 | 221 | 0 | 0 | 188
  Men W, Day 31 (Post vaccination) | 89.9 [61.9 to 130.7] | 122.6 [84.1 to 178.6] |  |  | 87.0 [59.0 to 128.3]
  Men W, Day 211 (Post vaccination): number analyzed (Participants) | 204 | 213 | 161 | 169 | 0
  Men W, Day 211 (Post vaccination) | 683.2 [572.6 to 815.1] | 800.6 [671.8 to 954.1] | 366.4 [303.4 to 442.5] | 481.0 [398.2 to 580.9] |
  Men Y, Day 1: number analyzed (Participants) | 207 | 211 | 0 | 0 | 193
  Men Y, Day 1 | 7.4 [6.3 to 8.7] | 7.7 [6.5 to 9.0] |  |  | 8.7 [7.4 to 10.3]
  Men Y, Day 31 (Pre vaccination): number analyzed (Participants) | 0 | 0 | 175 | 187 | 0
  Men Y, Day 31 (Pre vaccination) |  |  | 8.8 [7.4 to 10.4] | 7.7 [6.5 to 9.1] |
  Men Y, Day 31 (Post vaccination): number analyzed (Participants) | 222 | 226 | 0 | 0 | 190
  Men Y, Day 31 (Post vaccination) | 62.8 [43.8 to 90.2] | 64.2 [44.7 to 92.2] |  |  | 100.0 [68.7 to 145.5]
  Men Y, Day 211(Post vaccination): number analyzed (Participants) | 203 | 214 | 161 | 169 | 0
  Men Y, Day 211(Post vaccination) | 406.9 [315.8 to 524.4] | 353.1 [274.6 to 454.0] | 239.5 [182.7 to 314.0] | 215.1 [164.1 to 281.9] |

45. Secondary Outcome: hSBA GMRs Against Serogroups A, C, W and Y in Study Phase II (Formulation and Schedule-finding)
Description: For each serogroup A, C, W and Y, the GMRs (post-vaccination/ Day 1 (Month 0)) are calculated with their associated 2-sided 95% CIs, by exponentiating the corresponding log-transformed means and their 95% CIs.
Time Frame: At Day 31 [for ABCWY (0,6-months) and Control group compared to Day 1 (Baseline)], at Day 211 [for ABCWY (0,6-months) groups compared to Day 1 (baseline) and for ABCWY (0,2-months) groups compared to Day 31]
Population: as for outcome 37
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | ABCWY Low dose_06 Group | ABCWY High dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_02 Group | Control Group
Number analyzed (Participants) | 194 | 201 | 159 | 171 | 186
Ratio
  Men A, Day 31: number analyzed (Participants) | 176 | 186 | 0 | 0 | 180
  Men A, Day 31 | 19.1 [14.2 to 25.8] | 17.0 [12.5 to 22.9] |  |  | 42.9 [31.9 to 57.8]
  Men A, Day 211: number analyzed (Participants) | 177 | 181 | 152 | 163 | 0
  Men A, Day 211 | 43.0 [35.3 to 52.5] | 53.3 [43.6 to 65.3] | 38.4 [31.2 to 47.4] | 45.8 [37.3 to 56.3] |
  Men C, Day 31: number analyzed (Participants) | 193 | 192 | 0 | 0 | 178
  Men C, Day 31 | 14.8 [9.6 to 22.7] | 13.9 [8.9 to 21.6] |  |  | 15.6 [10.0 to 24.2]
  Men C, Day 211: number analyzed (Participants) | 180 | 190 | 156 | 171 | 0
  Men C, Day 211 | 91.5 [68.4 to 122.5] | 78.4 [58.5 to 105.1] | 77.3 [57.0 to 104.8] | 66.2 [49.1 to 89.4] |
  Men W, Day 31: number analyzed (Participants) | 194 | 195 | 0 | 0 | 183
  Men W, Day 31 | 13.2 [9.3 to 18.8] | 17.5 [12.2 to 24.9] |  |  | 12.5 [8.7 to 17.9]
  Men W, Day 211: number analyzed (Participants) | 178 | 189 | 157 | 167 | 0
  Men W, Day 211 | 101.6 [78.7 to 131.2] | 127.9 [99.4 to 164.7] | 54.0 [41.4 to 70.4] | 69.8 [53.6 to 90.9] |
  Men Y, Day 31: number analyzed (Participants) | 193 | 201 | 0 | 0 | 186
  Men Y, Day 31 | 9.5 [6.6 to 13.7] | 9.3 [6.4 to 13.4] |  |  | 13.1 [9.0 to 19.0]
  Men Y, Day 211: number analyzed (Participants) | 177 | 192 | 159 | 167 | 0
  Men Y, Day 211 | 61.6 [46.3 to 81.8] | 51.7 [39.0 to 68.4] | 32.2 [24.0 to 43.2] | 31.6 [23.5 to 42.3] |

46. Secondary Outcome: Immunoglobulin G (IgG) Antibodies Against Serogroups A, C, W and Y in Study Phase II (Formulation and Schedule-finding)
Description: The immune responses to MenABCWY-2Gen (low and high dose) and MenACWY vaccines are evaluated by measuring the total IgG in terms of electrochemiluminescence-based (ECL) multiplex assay Geometric Mean Concentrations (GMCs).
Time Frame: as for outcome 42
Population: as for outcome 37
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram per milliliter(µg/mL)
Arm/Group | ABCWY Low dose_06 Group | ABCWY High dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_02 Group | Control Group
Number analyzed (Participants) | 211 | 223 | 170 | 184 | 187
Microgram per milliliter(µg/mL)
  Men A Ab, Day 1: number analyzed (Participants) | 197 | 201 | 0 | 0 | 176
  Men A Ab, Day 1 | 2.3 [2.0 to 2.6] | 2.1 [1.8 to 2.4] |  |  | 2.3 [2.0 to 2.6]
  Men A Ab, Day 31 (Pre vaccination): number analyzed (Participants) | 0 | 0 | 168 | 184 | 0
  Men A Ab, Day 31 (Pre vaccination) |  |  | 2.4 [2.1 to 2.8] | 2.3 [2.0 to 2.7] |
  Men A Ab, Day 31 (Post vaccination): number analyzed (Participants) | 207 | 221 | 0 | 0 | 183
  Men A Ab, Day 31 (Post vaccination) | 10.5 [8.0 to 13.8] | 9.3 [7.1 to 12.2] |  |  | 20.3 [15.4 to 26.7]
  Men A Ab, Day 211 (Post vaccination): number analyzed (Participants) | 178 | 189 | 135 | 139 | 0
  Men A Ab, Day 211 (Post vaccination) | 14.6 [11.5 to 18.6] | 13.1 [10.4 to 16.5] | 14.0 [10.9 to 18.1] | 14.0 [10.9 to 18.1] |
  Men C Ab, Day 1: number analyzed (Participants) | 197 | 202 | 0 | 0 | 178
  Men C Ab, Day 1 | 1.1 [1.0 to 1.2] | 1.1 [1.0 to 1.2] |  |  | 1.1 [1.0 to 1.3]
  Men C Ab, Day 31 (Pre vaccination): number analyzed (Participants) | 0 | 0 | 169 | 183 | 0
  Men C Ab, Day 31 (Pre vaccination) |  |  | 1.0 [0.9 to 1.1] | 1.1 [1.0 to 1.2] |
  Men C Ab, Day 31 (Post vaccination): number analyzed (Participants) | 208 | 217 | 0 | 0 | 181
  Men C Ab, Day 31 (Post vaccination) | 8.0 [6.1 to 10.6] | 8.1 [6.2 to 10.7] |  |  | 8.6 [6.5 to 11.4]
  Men C Ab, Day 211 (Post vaccination): number analyzed (Participants) | 164 | 172 | 116 | 128 | 0
  Men C Ab, Day 211 (Post vaccination) | 8.6 [6.9 to 10.7] | 8.0 [6.5 to 9.8] | 11.7 [9.3 to 14.8] | 11.2 [8.9 to 14.1] |
  Men W Ab, Day 1: number analyzed (Participants) | 197 | 201 | 0 | 0 | 178
  Men W Ab, Day 1 | 1.3 [1.1 to 1.4] | 1.2 [1.1 to 1.3] |  |  | 1.2 [1.1 to 1.4]
  Men W Ab, Day 31 (Pre vaccination): number analyzed (Participants) | 0 | 0 | 170 | 182 | 0
  Men W Ab, Day 31 (Pre vaccination) |  |  | 1.2 [1.1 to 1.4] | 1.2 [1.1 to 1.4] |
  Men W Ab, Day 31 (Post vaccination): number analyzed (Participants) | 211 | 223 | 0 | 0 | 187
  Men W Ab, Day 31 (Post vaccination) | 4.6 [3.5 to 6.1] | 4.3 [3.3 to 5.7] |  |  | 3.6 [2.7 to 4.8]
  Men W Ab, Day 211 (Post vaccination): number analyzed (Participants) | 180 | 187 | 125 | 136 | 0
  Men W Ab, Day 211 (Post vaccination) | 8.2 [6.4 to 10.5] | 8.7 [6.8 to 11.1] | 6.2 [4.7 to 8.1] | 7.2 [5.5 to 9.5] |
  Men Y Ab, Day 1: number analyzed (Participants) | 196 | 202 | 0 | 0 | 177
  Men Y Ab, Day 1 | 1.3 [1.2 to 1.5] | 1.3 [1.2 to 1.4] |  |  | 1.3 [1.2 to 1.5]
  Men Y Ab, Day 31 (Pre vaccination): number analyzed (Participants) | 0 | 0 | 169 | 183 | 0
  Men Y Ab, Day 31 (Pre vaccination) |  |  | 1.4 [1.2 to 1.5] | 1.3 [1.2 to 1.4] |
  Men Y Ab, Day 31 (Post vaccination): number analyzed (Participants) | 208 | 221 | 0 | 0 | 185
  Men Y Ab, Day 31 (Post vaccination) | 4.2 [3.2 to 5.5] | 4.4 [3.4 to 5.8] |  |  | 5.3 [4.0 to 7.0]
  Men Y Ab, Day 211 (Post vaccination): number analyzed (Participants) | 180 | 189 | 136 | 139 | 0
  Men Y Ab, Day 211 (Post vaccination) | 10.1 [7.8 to 13.1] | 10.0 [7.8 to 12.9] | 11.3 [8.6 to 15.0] | 9.8 [7.4 to 12.9] |

ADVERSE EVENTS:
Time Frame: Solicited AEs: during the 7-day follow-up period after any vaccination and Unsolicited AEs: during the 30-day follow-up period after any vaccination in all the 3 phases. SAEs, AEs leading to withdrawal & AESIs were collected throughout the study period: from Day 1 up to study end [Day 211] in Phase I (Safety Lead-in); from Day 1 up to study end [Day 541] in Phase II (Formulation and Schedule-Finding); from Day 1 up to study end [Day 361] in Phase II (Sourcing).
Arm/Group | ABCWY Low Dose Group | Placebo Low Dose Group | ABCWY High Dose Group | Placebo High Dose Group | ABCWY Low dose_06 Group | ABCWY Low dose_02 Group | ABCWY High dose_06 Group | ABCWY High dose_02 Group | Control Group | ABCWY Low dose_01 Group | ABCWY High dose_01 Group | ABCWY Low doseS_02 Group | ABCWY High doseS_02 Group | ABCWY Low doseS_06 Group | ABCWY High doseS_06 Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/4 | 0/13 | 0/3 | 0/239 | 0/181 | 0/238 | 0/194 | 0/197 | 0/54 | 0/53 | 0/62 | 0/62 | 0/62 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/4 | 0/13 | 0/3 | 9/239 | 7/181 | 4/238 | 4/194 | 2/197 | 0/54 | 0/53 | 2/62 | 1/62 | 0/62 | 4/63
Other Adverse Events (participants affected / at risk) | 12/12 | 3/4 | 13/13 | 2/3 | 229/239 | 170/181 | 234/238 | 182/194 | 192/197 | 50/54 | 53/53 | 61/62 | 58/62 | 60/62 | 62/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABCWY Low Dose Group (N=12) | Placebo Low Dose Group (N=4) | ABCWY High Dose Group (N=13) | Placebo High Dose Group (N=3) | ABCWY Low dose_06 Group (N=239) | ABCWY Low dose_02 Group (N=181) | ABCWY High dose_06 Group (N=238) | ABCWY High dose_02 Group (N=194) | Control Group (N=197) | ABCWY Low dose_01 Group (N=54) | ABCWY High dose_01 Group (N=53) | ABCWY Low doseS_02 Group (N=62) | ABCWY High doseS_02 Group (N=62) | ABCWY Low doseS_06 Group (N=62) | ABCWY High doseS_06 Group (N=63)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mesenteric lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign familial haematuria (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterobiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pilonidal disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bell's palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranoid personality disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABCWY Low Dose Group (N=12) | Placebo Low Dose Group (N=4) | ABCWY High Dose Group (N=13) | Placebo High Dose Group (N=3) | ABCWY Low dose_06 Group (N=239) | ABCWY Low dose_02 Group (N=181) | ABCWY High dose_06 Group (N=238) | ABCWY High dose_02 Group (N=194) | Control Group (N=197) | ABCWY Low dose_01 Group (N=54) | ABCWY High dose_01 Group (N=53) | ABCWY Low doseS_02 Group (N=62) | ABCWY High doseS_02 Group (N=62) | ABCWY Low doseS_06 Group (N=62) | ABCWY High doseS_06 Group (N=63)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inner ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperprolactinaemia (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polycystic ovarian syndrome (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panophthalmitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 4 (5) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 2 (2) | 6 (6) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (2) | 4 (5) | 0 (0) | 57 (68) | 34 (37) | 57 (69) | 35 (47) | 30 (35) | 9 (11) | 13 (15) | 10 (12) | 10 (11) | 11 (12) | 11 (14)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Administration site erythema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 46 (56) | 25 (33) | 45 (51) | 29 (32) | 32 (37) | 14 (16) | 8 (11) | 22 (33) | 20 (28) | 26 (31) | 24 (28)
Administration site hypoaesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Administration site induration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 32 (41) | 27 (34) | 44 (50) | 27 (35) | 29 (32) | 8 (9) | 9 (12) | 18 (26) | 18 (20) | 16 (21) | 20 (25)
Administration site pain (General disorders) | 11 (19) | 2 (2) | 13 (21) | 1 (1) | 226 (443) | 160 (321) | 232 (440) | 173 (346) | 186 (340) | 50 (91) | 51 (86) | 61 (110) | 55 (98) | 59 (107) | 60 (102)
Administration site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 48 (62) | 34 (47) | 52 (59) | 33 (45) | 31 (35) | 10 (11) | 14 (22) | 25 (36) | 22 (28) | 24 (31) | 26 (34)
Administration site warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 6 (7) | 3 (3) | 12 (18) | 2 (4) | 152 (256) | 104 (193) | 147 (252) | 115 (206) | 118 (167) | 31 (45) | 36 (51) | 50 (78) | 37 (51) | 49 (71) | 41 (56)
Hangover (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 8 (14) | 12 (17) | 8 (14) | 5 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site hypoaesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site lymphadenopathy (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 2 (5) | 0 (0) | 5 (5) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site paraesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 14 (15) | 12 (13) | 18 (21) | 10 (10) | 15 (16) | 3 (3) | 7 (7) | 3 (3) | 3 (3) | 5 (5) | 5 (5)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaccination site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaccination site warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mite allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mycotic allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alveolar osteitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 14 (14) | 14 (16) | 12 (12) | 16 (17) | 6 (6) | 4 (4) | 5 (5) | 3 (3) | 4 (4) | 2 (2) | 3 (3)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chlamydial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (10) | 4 (4) | 7 (7) | 7 (7) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lyme disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 21 (26) | 14 (18) | 17 (22) | 12 (15) | 5 (5) | 0 (0) | 0 (0) | 3 (3) | 2 (3) | 4 (4) | 4 (5)
Norovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 3 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pharyngitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post-acute COVID-19 syndrome (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pustule (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 5 (7) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 3 (3) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 16 (19) | 8 (11) | 12 (15) | 8 (8) | 12 (12) | 2 (2) | 2 (2) | 1 (2) | 4 (5) | 2 (2) | 7 (7)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral rash (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vulval abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heat exhaustion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immunisation reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Repetitive strain injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Human metapneumovirus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Streptococcus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypovitaminosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insulin resistance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 4 (4) | 1 (1) | 27 (33) | 26 (29) | 44 (51) | 21 (27) | 20 (21) | 10 (11) | 11 (15) | 11 (15) | 13 (14) | 15 (20) | 20 (29)
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaw disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1) | 6 (7) | 1 (1) | 53 (63) | 34 (45) | 57 (71) | 41 (55) | 47 (51) | 18 (21) | 18 (25) | 19 (23) | 17 (20) | 25 (27) | 23 (30)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 7 (11) | 2 (2) | 5 (9) | 2 (2) | 140 (234) | 110 (180) | 157 (250) | 112 (190) | 104 (146) | 33 (43) | 29 (41) | 38 (52) | 31 (44) | 36 (49) | 37 (47)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine with aura (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anger (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Eating disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Initial insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obsessive-compulsive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Social anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urethral pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Menstrual disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 4 (4) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (8) | 6 (7) | 7 (7) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (6) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychalgia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parapsoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sea bather's eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria chronic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/54/NCT04886154/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-29): https://cdn.clinicaltrials.gov/large-docs/54/NCT04886154/SAP_001.pdf